CLINICAL TRIAL: NCT04493684
Title: A Double-Blind (Sponsor Unblinded), Randomized, Placebo-Controlled, Single and Repeated Dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics of GSK3739937 in Healthy Participants
Brief Title: GSK3739937 First-Time-In-Human (FTIH) Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 212548
Record Dates: First submitted 2020-07-20; First posted 2020-07-30 (Actual); Results first posted 2023-08-23 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; First-time-in-human; Pharmacokinetics; Safety; Tolerability
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Tablets

STUDY DESIGN:
Intervention Model Description: Part 1 is a single ascending dose study, Part 2 is multiple ascending dose study while Part 3 is a 3-period crossover design.
Who Masked: Participant, Investigator
Masking Description: This will be a double-blind study with participants and the site-staff blinded and sponsor unblended. Part 3 of the study will be open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Part 1: Cohort 1: Participants receiving GSK3739937 (Experimental): Part 1 cohort 1 may contain up to 4 escalating doses (Period 1- 10 milligram [mg], Period 2- 80 mg, and Period 3- 320 mg, Period 4- 800 mg) of GSK3739937.
  Interventions: Drug: GSK3739937 (PIB)
- Part 1: Cohort 1: Participants receiving Placebo (Placebo Comparator): In this cohort, participants will be randomized to receive placebo.
  Interventions: Drug: Placebo
- Part 1: Cohort 2: Participants receiving GSK3739937 (Experimental): Part 1 cohort 2 may contain up to 3 escalating doses ( Period 1- 30 mg, Period 2- 160 mg, and Period 3- 640 mg) of GSK3739937.
  Interventions: Drug: GSK3739937 (PIB)
- Part 1: Cohort 2: Participants receiving Placebo (Placebo Comparator): In this cohort, participants will be randomized to receive placebo.
  Interventions: Drug: Placebo
- Part 2: Cohort 3: Participants receiving GSK3739937 (Experimental): Eligible participants in part 2 cohort 3, will consist of approximately 10 participants out of 7 participants will be randomized to receive a once-daily dose of 25 mg GSK3739937 for 14 days.
  Interventions: Drug: GSK3739937 (PIB)
- Part 2: Cohort 3: Participants receiving Placebo (Placebo Comparator): Eligible participants in part 2 cohort 3, will consist of approximately 10 participants out of 3 participants will be randomized to receive a once-daily dose of placebo for 14 days.
  Interventions: Drug: Placebo
- Part 2: Cohort 4: Participants receiving GSK3739937 (Experimental): Eligible participants in part 2 cohort 4, will consist of approximately 10 participants out of 7 participants will be randomized to receive a once-daily dose of 50 mg GSK3739937 for 14 days.
  Interventions: Drug: GSK3739937 (PIB)
- Part 2: Cohort 4: Participants receiving Placebo (Placebo Comparator): Eligible participants in part 2 cohort 4, will consist of approximately 10 participants out of 3 participants will be randomized to receive a once-daily dose of placebo for 14 days.
  Interventions: Drug: Placebo
- Part 2: Cohort 5: Participants receiving GSK3739937 (Experimental): Eligible participants in part 2 cohort 5, will consist of approximately 10 participants out of 7 participants will be randomized to receive a once-daily dose of 100 mg GSK3739937 for 18 days.
  Interventions: Drug: GSK3739937 (PIB)
- Part 2: Cohort 5: Participants receiving placebo (Placebo Comparator): Eligible participants in part 2 cohort 5, will consist of approximately 10 participants out of 3 participants will be randomized to receive a once-daily dose of placebo for 18 days.
  Interventions: Drug: Placebo
- Part 2: Cohort 6: Participants receiving GSK3739937 (Experimental): Eligible participants in part 2 cohort 6, will consist of approximately 10 participants out of 7 participants will be randomized to receive three 500 mg doses of GSK3739937 administered at once weekly intervals over two weeks.
  Interventions: Drug: GSK3739937 (PIB)
- Part 2: Cohort 6: Participants receiving placebo (Placebo Comparator): Eligible participants in part 2 cohort 6, will consist of approximately 10 participants out of 3 participants will be randomized to receive three doses of placebo administered at once weekly intervals over two weeks.
  Interventions: Drug: Placebo
- Part 3: Cohort 7: Participants receiving treatment sequence ABC (Experimental): Participants will receive Treatment A: GSK3739937 PiB, 100 mg administered under moderate fat conditions in Period 1; Treatment B: GSK3739937 Tablet, 100 mg administered under moderate fat conditions in Period 2; and Treatment C: GSK3739937 Tablet, 100 mg administered under fasted conditions in Period 3.
  Interventions: Drug: GSK3739937 (PIB); Drug: GSK3739937 (Tablet)
- Part 3: Cohort 7: Participants receiving treatment sequence BCA (Experimental): Participants will receive Treatment B: GSK3739937 Tablet, 100 mg administered under moderate fat conditions in Period 1; Treatment C: GSK3739937 Tablet, 100 mg administered under fasted conditions in Period 2; and Treatment A: GSK3739937 PiB, 100 mg administered under moderate fat conditions in Period 3.
  Interventions: Drug: GSK3739937 (PIB); Drug: GSK3739937 (Tablet)
- Part 3: Cohort 7: Participants receiving treatment sequence CAB (Experimental): Participants will receive Treatment C: GSK3739937 Tablet, 100 mg administered under fasted conditions in Period 1; Treatment A: GSK3739937 PiB, 100 mg administered under moderate fat conditions in Period 2; and Treatment B: GSK3739937 Tablet, 100 mg administered under moderate fat conditions in Period 3.
  Interventions: Drug: GSK3739937 (PIB); Drug: GSK3739937 (Tablet)

INTERVENTIONS:
Drug: GSK3739937 (PIB) — GSK3739937 will be administered as oral suspension.
  Arms: Part 1: Cohort 1: Participants receiving GSK3739937; Part 1: Cohort 2: Participants receiving GSK3739937; Part 2: Cohort 3: Participants receiving GSK3739937; Part 2: Cohort 4: Participants receiving GSK3739937; Part 2: Cohort 5: Participants receiving GSK3739937; Part 2: Cohort 6: Participants receiving GSK3739937; Part 3: Cohort 7: Participants receiving treatment sequence ABC; Part 3: Cohort 7: Participants receiving treatment sequence BCA; Part 3: Cohort 7: Participants receiving treatment sequence CAB
Drug: Placebo — Placebo will be given orally during each dosing day.
  Arms: Part 1: Cohort 1: Participants receiving Placebo; Part 1: Cohort 2: Participants receiving Placebo; Part 2: Cohort 3: Participants receiving Placebo; Part 2: Cohort 4: Participants receiving Placebo; Part 2: Cohort 5: Participants receiving placebo; Part 2: Cohort 6: Participants receiving placebo
Drug: GSK3739937 (Tablet) — GSK3739937 Tablet will be administered via oral route.
  Arms: Part 3: Cohort 7: Participants receiving treatment sequence ABC; Part 3: Cohort 7: Participants receiving treatment sequence BCA; Part 3: Cohort 7: Participants receiving treatment sequence CAB

SUMMARY:
This study is a Phase 1, double-blind (sponsor-unblinded), randomized, placebo-controlled, single- and repeat-dose escalation study including a weekly oral dose (MAD) cohort and a relative bioavailability (RBA) and food effect (FE) cohort to investigate the safety, tolerability and PK of VH3739937 in healthy participants. This is a three part study. Part 1 and Part 2 is designed to gain information on the safety, tolerability, and pharmacokinetic (PK) properties of GSK3739937 when administered as powder-in-a-bottle (PiB). Part 3 will evaluate the RBA of the GSK3739937 PiB and GSK3739937 Tablet and the safety, tolerability and PK parameters of the tablet formulation when administered under fasting and fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring (history and ECG).
* Participants who are negative on two consecutive tests for severe acute respiratory syndrome coronavirus-2 (SARs-CoV-2), performed at Screening and on admission and (re-)admission to the Phase I unit, using an approved molecular test polymerase chain reaction (PCR).
* Participants who are able to understand and comply with protocol requirements and timetables, instructions, and protocol-stated restrictions.
* Body weight >=50.0 kilograms (kg) (110 pound [lbs]) for men and >=45.0 kg (99 lbs) for women and body mass index within the range 18.5 to 32.0 kilogram per square meter (kg/m^2).
* Male participants are eligible to participate if they agree to use contraceptive methods
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and is not a woman of childbearing potential (WOCBP). - Capable of giving signed informed consent

Exclusion Criteria:

* Signs and symptoms which in the opinion of the investigator are suggestive of coronavirus disease 2019 (COVID-19) (i.e. fever, cough etc) within 14 days of inpatient admission.
* Contact with known COVID-19 positive persons in the 14 days prior to inpatient admission.
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, distribution, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
* Pre-existing clinically relevant, in the opinion of the principal investigator (PI), gastro-intestinal pathology or diagnosis - e.g. irritable bowel syndrome, inflammatory bowel disease, and/or significant baseline signs and symptoms.
* Medical history of cardiac arrhythmias or cardiac disease or a family and personal history of long QT syndrome.
* Any known or suspected pre-existing psychiatric condition
* Any positive (abnormal) response confirmed by the investigator or clinician (or qualified designee) administered Columbia Suicide Severity Rating Scale (CSSRS) at screening .
* Any other clinical condition (including but not limited to active substance use) or prior therapy that, in the opinion of the Investigator, would make the participant unsuitable for the study; unable to comply with dosing requirements; or unable to comply with study visits; or a condition that could affect the absorption, distribution, metabolism or excretion of the drug.
* Estimated glomerular filtration rate (eGFR) <90 milliliters/minute (mL/min) or serum creatinine >1.1 x upper limit of normal (ULN).
* Hemoglobin <12.5 grams/deciliter (g/dL) for men and <11 g/dL for women.
* ALT or AST >1.1x ULN.
* Bilirubin >1.1 x ULN (isolated bilirubin >1.1 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Any significant arrhythmia or ECG finding (e.g., prior myocardial infarction in the past 3 months (does not include ST segment changes associated with repolarization), symptomatic bradycardia, non-sustained or sustained atrial arrhythmias, non-sustained or sustained ventricular tachycardia (>=3 consecutive ventricular ectopic beats), second-degree atrioventricular (AV) block Mobitz Type II, third-degree atrioventricular block, complete heart block, or conduction abnormality (including but not specific to left or right complete bundle branch; AV block [2nd degree or higher]; Wolff-Parkinson-White [WPW] syndrome), Sinus Pauses > 3 seconds, which, in the opinion of the investigator or ViiV Healthcare (VH)/ GlaxoSmithKline (GSK) Medical Monitor, will interfere with the safety for the individual participant.
* Exclusion criteria for Screening ECG. Heart rate <45 or >100 beats per minute (bpm) for males and <50 or >100 bpm for females; PR interval <120 or >220 millisecond (msec); QRS duration <70 or >120 msec; the Fridericia's QT correction formula (QTcF) interval >450 msec.
* Past or intended use of over-the-counter or prescription medication [including cytochrome p450 enzyme inducers or inhibitors, vitamins, herbal and dietary supplements ] within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to dosing and for the duration of the study, unless in the opinion of the Investigator and Sponsor, the medication will not interfere with the study medications, procedures, or compromise participant safety.
* Unwillingness to abstain from ingestion of any food or drink containing grapefruit and grapefruit juice, Seville oranges, blood oranges, or pomelos within 7 days prior to the first dose of study treatments or until the end of the study.
* Participation in the study would result in loss of blood or blood products in excess of 500 mL within 56 days
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day
* Current enrolment or past participation within the last 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) before signing of consent in this or any other clinical study involving an investigational study intervention or any other type of medical research
* Presence of Hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study intervention
* Positive Hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
* Positive Hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention
* Positive pre-study drug/alcohol screen
* Positive HIV antibody/antigen test
* Regular use of known drugs of abuse
* Regular alcohol consumption within 6 months prior to the study defined as: An average weekly intake of >14 units for males or >7 units for females.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products (e.g. nicotine patches or vaporizing devices) within 6 months prior to screening and at admission.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/en/study/?id=212548
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf

REFERENCES:
- [Background] Benn PD, Zhang Y, Kahl L, Greene TJ, Bainbridge V, Fishman C, Wen B, Gartland M. A phase I, first-in-human study investigating the safety, tolerability, and pharmacokinetics of the maturation inhibitor GSK3739937. Pharmacol Res Perspect. 2023 Jun;11(3):e01093. doi: 10.1002/prp2.1093. PMID 37269076

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study includes 3 parts. In part 1, 34 participants were randomized. In part 2, 40 participants were randomized. In part 3, 17 participants were randomized.
Groups:
- Part 1 (Cohort 1) - Single Dose (SD) Placebo (PBO)/GSK3739937 SD 80 mg/GSK3739937 SD 320 mg: Participants received single oral dose of placebo as suspension in Treatment Period 1, followed by single oral dose of 80 milligrams (mg) of GSK3739937 in Treatment Period 2, and followed by single oral dose of 320 mg of GSK3739937 in Treatment Period 3.
- Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ SD PBO/ GSK3739937 SD 320 mg: Participants received single oral dose of 10 mg of GSK3739937 as suspension in Treatment Period 1, followed by single oral dose of placebo as suspension in Treatment Period 2, and followed by single oral dose of 320 mg of GSK3739937 as suspension in Treatment Period 3.
- Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ GSK3739937 SD 80 mg/SD PBO: Participants received single oral dose of 10 mg of GSK3739937 as suspension in Treatment Period 1, followed by single oral dose of 80 mg of GSK3739937 as suspension in Treatment Period 2, and followed by single oral dose of placebo as suspension in Treatment Period 3.
- Part 1 (Cohort 1) - GSK3739937 SD 800 mg: Participants received single oral dose of 800 mg of GSK3739937 as suspension in Treatment Period 1.
- Part 1 (Cohort 1) - SD PBO: Participants received single oral dose of Placebo in Treatment Period 1.
- Part 1 (Cohort 2) - SD PBO/ GSK3739937 SD 160 mg/ GSK3739937 SD 640 mg: Participants received single oral dose of Placebo as suspension in Treatment Period 1, followed by single oral dose of 160 mg of GSK3739937 as suspension in Treatment Period 2, and followed by single oral dose of 640 mg of GSK3739937 as suspension Treatment in Period 3.
- Part 1 (Cohort 2) - GSK3739937 SD 30mg/ SD PBO/ GSK3739937 SD 640mg: Participants received single oral dose of 30 mg of GSK3739937 as suspension in Treatment Period 1, followed by single oral dose of Placebo as suspension in Treatment Period 2, and followed by single oral dose of 640 mg of GSK3739937 as suspension in Treatment Period 3.
- Part 1 (Cohort 2) - GSK3739937 SD 30 mg/ GSK3739937 SD 160 mg/SD PBO: Participants received single oral dose of 30 mg of GSK3739937 as suspension in Treatment Period 1, followed by single oral dose of 160 mg of GSK3739937 in Period 2, and followed by single oral dose of Placebo in Period 3.
- Part 2 - Once Daily (QD) PBO: Participants received once daily oral doses of Placebo as suspension for 14 days in Treatment Period 1.
- Part 2 (Cohort 3) - GSK3739937 QD 25 mg: Participants received once daily oral doses of 25 mg of GSK3739937 as suspension for 14 days in Treatment Period 1.
- Part 2 (Cohort 4) - GSK3739937 QD 50 mg: Participants received once daily oral doses of 50 mg of GSK3739937 as suspension for 14 days in Treatment Period 1.
- Part 2 (Cohort 5) - GSK3739937 QD 100 mg: Participants received once daily oral doses of 100 mg of GSK3739937 as suspension for 18 days in Treatment Period 1.
- Part 2 - Once Weekly (QW) PBO: Participants received once weekly oral doses of Placebo as suspension for over 3 weeks in Treatment Period 1.
- Part 2 (Cohort 6) - GSK3739937 QW 500 mg: Participants received once weekly oral doses of 500 mg of GSK3739937 as suspension for over 3 weeks in Treatment Period 1.
- Part 3 (Cohort 7) - GSK3739937 PiB Fed/ GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted: Participants received single dose of 100 mg of powder in bottle (PiB) as oral suspension under moderate fed conditions in Treatment Period 1, followed by single oral dose of 100 mg of GSK3739937 tablet under moderate fed conditions in Treatment Period 2 and followed by single dose of 100 mg of GSK3739937 tablet under fasted conditions in Treatment Period 3.
- Part 3 (Cohort 7) - GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed: Participants received single oral dose of 100 mg of GSK3739937 tablet under moderate fed conditions in Treatment Period 1, followed by single oral dose of 100 mg GSK3739937 tablet under fasted conditions in Treatment Period 2 and followed by single dose of 100 mg PiB as oral suspension under moderate fed conditions in Treatment Period 3.
- Part 3 (Cohort 7) - GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed/ GSK3739937 Tablet Fed: Participants received single oral dose of 100 mg of GSK3739937 tablet under fasted condition in Treatment Period 1, followed by single oral dose of 100 mg PiB as oral suspension under moderate fed conditions in Treatment Period 2 and followed by single oral dose of 100 mg GSK3739937 tablet under fed conditions in Treatment Period 3.
Period: Part 1:Treatment Period 1-Up to 9 Weeks
Arm/Group | Part 1 (Cohort 1) - Single Dose (SD) Placebo (PBO)/GSK3739937 SD 80 mg/GSK3739937 SD 320 mg | Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ SD PBO/ GSK3739937 SD 320 mg | Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ GSK3739937 SD 80 mg/SD PBO | Part 1 (Cohort 1) - GSK3739937 SD 800 mg | Part 1 (Cohort 1) - SD PBO | Part 1 (Cohort 2) - SD PBO/ GSK3739937 SD 160 mg/ GSK3739937 SD 640 mg | Part 1 (Cohort 2) - GSK3739937 SD 30mg/ SD PBO/ GSK3739937 SD 640mg | Part 1 (Cohort 2) - GSK3739937 SD 30 mg/ GSK3739937 SD 160 mg/SD PBO | Part 2 - Once Daily (QD) PBO | Part 2 (Cohort 3) - GSK3739937 QD 25 mg | Part 2 (Cohort 4) - GSK3739937 QD 50 mg | Part 2 (Cohort 5) - GSK3739937 QD 100 mg | Part 2 - Once Weekly (QW) PBO | Part 2 (Cohort 6) - GSK3739937 QW 500 mg | Part 3 (Cohort 7) - GSK3739937 PiB Fed/ GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted | Part 3 (Cohort 7) - GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed | Part 3 (Cohort 7) - GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed/ GSK3739937 Tablet Fed
Started | 3 | 3 | 3 | 6 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 3 | 2 | 6 | 3 | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1:Treatment Period 2-Up to 9 Weeks
Arm/Group | Part 1 (Cohort 1) - Single Dose (SD) Placebo (PBO)/GSK3739937 SD 80 mg/GSK3739937 SD 320 mg | Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ SD PBO/ GSK3739937 SD 320 mg | Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ GSK3739937 SD 80 mg/SD PBO | Part 1 (Cohort 1) - GSK3739937 SD 800 mg | Part 1 (Cohort 1) - SD PBO | Part 1 (Cohort 2) - SD PBO/ GSK3739937 SD 160 mg/ GSK3739937 SD 640 mg | Part 1 (Cohort 2) - GSK3739937 SD 30mg/ SD PBO/ GSK3739937 SD 640mg | Part 1 (Cohort 2) - GSK3739937 SD 30 mg/ GSK3739937 SD 160 mg/SD PBO | Part 2 - Once Daily (QD) PBO | Part 2 (Cohort 3) - GSK3739937 QD 25 mg | Part 2 (Cohort 4) - GSK3739937 QD 50 mg | Part 2 (Cohort 5) - GSK3739937 QD 100 mg | Part 2 - Once Weekly (QW) PBO | Part 2 (Cohort 6) - GSK3739937 QW 500 mg | Part 3 (Cohort 7) - GSK3739937 PiB Fed/ GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted | Part 3 (Cohort 7) - GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed | Part 3 (Cohort 7) - GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed/ GSK3739937 Tablet Fed
Started | 4 (2 additional participants were enrolled and dosed.) | 3 | 3 (1 additional participant was enrolled and dosed.) | 0 | 0 | 3 (1 additional participant was enrolled and dosed.) | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 0 | 0 | 3 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1:Treatment Period 3-Up to 9 Weeks
Arm/Group | Part 1 (Cohort 1) - Single Dose (SD) Placebo (PBO)/GSK3739937 SD 80 mg/GSK3739937 SD 320 mg | Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ SD PBO/ GSK3739937 SD 320 mg | Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ GSK3739937 SD 80 mg/SD PBO | Part 1 (Cohort 1) - GSK3739937 SD 800 mg | Part 1 (Cohort 1) - SD PBO | Part 1 (Cohort 2) - SD PBO/ GSK3739937 SD 160 mg/ GSK3739937 SD 640 mg | Part 1 (Cohort 2) - GSK3739937 SD 30mg/ SD PBO/ GSK3739937 SD 640mg | Part 1 (Cohort 2) - GSK3739937 SD 30 mg/ GSK3739937 SD 160 mg/SD PBO | Part 2 - Once Daily (QD) PBO | Part 2 (Cohort 3) - GSK3739937 QD 25 mg | Part 2 (Cohort 4) - GSK3739937 QD 50 mg | Part 2 (Cohort 5) - GSK3739937 QD 100 mg | Part 2 - Once Weekly (QW) PBO | Part 2 (Cohort 6) - GSK3739937 QW 500 mg | Part 3 (Cohort 7) - GSK3739937 PiB Fed/ GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted | Part 3 (Cohort 7) - GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed | Part 3 (Cohort 7) - GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed/ GSK3739937 Tablet Fed
Started | 4 (1 additional participant was enrolled and dosed.) | 3 | 3 | 0 | 0 | 4 (1 additional participant was enrolled and dosed.) | 3 (1 additional participant was enrolled and dosed.) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 0 | 0 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2:Treatment Period 1-Up to 5 Weeks
Arm/Group | Part 1 (Cohort 1) - Single Dose (SD) Placebo (PBO)/GSK3739937 SD 80 mg/GSK3739937 SD 320 mg | Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ SD PBO/ GSK3739937 SD 320 mg | Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ GSK3739937 SD 80 mg/SD PBO | Part 1 (Cohort 1) - GSK3739937 SD 800 mg | Part 1 (Cohort 1) - SD PBO | Part 1 (Cohort 2) - SD PBO/ GSK3739937 SD 160 mg/ GSK3739937 SD 640 mg | Part 1 (Cohort 2) - GSK3739937 SD 30mg/ SD PBO/ GSK3739937 SD 640mg | Part 1 (Cohort 2) - GSK3739937 SD 30 mg/ GSK3739937 SD 160 mg/SD PBO | Part 2 - Once Daily (QD) PBO | Part 2 (Cohort 3) - GSK3739937 QD 25 mg | Part 2 (Cohort 4) - GSK3739937 QD 50 mg | Part 2 (Cohort 5) - GSK3739937 QD 100 mg | Part 2 - Once Weekly (QW) PBO | Part 2 (Cohort 6) - GSK3739937 QW 500 mg | Part 3 (Cohort 7) - GSK3739937 PiB Fed/ GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted | Part 3 (Cohort 7) - GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed | Part 3 (Cohort 7) - GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed/ GSK3739937 Tablet Fed
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 7 | 7 | 7 | 3 | 7 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 7 | 7 | 6 | 3 | 7 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part 3:Treatment Period 1-Up to 4 Weeks
Arm/Group | Part 1 (Cohort 1) - Single Dose (SD) Placebo (PBO)/GSK3739937 SD 80 mg/GSK3739937 SD 320 mg | Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ SD PBO/ GSK3739937 SD 320 mg | Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ GSK3739937 SD 80 mg/SD PBO | Part 1 (Cohort 1) - GSK3739937 SD 800 mg | Part 1 (Cohort 1) - SD PBO | Part 1 (Cohort 2) - SD PBO/ GSK3739937 SD 160 mg/ GSK3739937 SD 640 mg | Part 1 (Cohort 2) - GSK3739937 SD 30mg/ SD PBO/ GSK3739937 SD 640mg | Part 1 (Cohort 2) - GSK3739937 SD 30 mg/ GSK3739937 SD 160 mg/SD PBO | Part 2 - Once Daily (QD) PBO | Part 2 (Cohort 3) - GSK3739937 QD 25 mg | Part 2 (Cohort 4) - GSK3739937 QD 50 mg | Part 2 (Cohort 5) - GSK3739937 QD 100 mg | Part 2 - Once Weekly (QW) PBO | Part 2 (Cohort 6) - GSK3739937 QW 500 mg | Part 3 (Cohort 7) - GSK3739937 PiB Fed/ GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted | Part 3 (Cohort 7) - GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed | Part 3 (Cohort 7) - GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed/ GSK3739937 Tablet Fed
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Part 3:Treatment Period 2-Up to 4 Weeks
Arm/Group | Part 1 (Cohort 1) - Single Dose (SD) Placebo (PBO)/GSK3739937 SD 80 mg/GSK3739937 SD 320 mg | Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ SD PBO/ GSK3739937 SD 320 mg | Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ GSK3739937 SD 80 mg/SD PBO | Part 1 (Cohort 1) - GSK3739937 SD 800 mg | Part 1 (Cohort 1) - SD PBO | Part 1 (Cohort 2) - SD PBO/ GSK3739937 SD 160 mg/ GSK3739937 SD 640 mg | Part 1 (Cohort 2) - GSK3739937 SD 30mg/ SD PBO/ GSK3739937 SD 640mg | Part 1 (Cohort 2) - GSK3739937 SD 30 mg/ GSK3739937 SD 160 mg/SD PBO | Part 2 - Once Daily (QD) PBO | Part 2 (Cohort 3) - GSK3739937 QD 25 mg | Part 2 (Cohort 4) - GSK3739937 QD 50 mg | Part 2 (Cohort 5) - GSK3739937 QD 100 mg | Part 2 - Once Weekly (QW) PBO | Part 2 (Cohort 6) - GSK3739937 QW 500 mg | Part 3 (Cohort 7) - GSK3739937 PiB Fed/ GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted | Part 3 (Cohort 7) - GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed | Part 3 (Cohort 7) - GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed/ GSK3739937 Tablet Fed
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Part 3:Treatment Period 3-Up to 4 Weeks
Arm/Group | Part 1 (Cohort 1) - Single Dose (SD) Placebo (PBO)/GSK3739937 SD 80 mg/GSK3739937 SD 320 mg | Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ SD PBO/ GSK3739937 SD 320 mg | Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ GSK3739937 SD 80 mg/SD PBO | Part 1 (Cohort 1) - GSK3739937 SD 800 mg | Part 1 (Cohort 1) - SD PBO | Part 1 (Cohort 2) - SD PBO/ GSK3739937 SD 160 mg/ GSK3739937 SD 640 mg | Part 1 (Cohort 2) - GSK3739937 SD 30mg/ SD PBO/ GSK3739937 SD 640mg | Part 1 (Cohort 2) - GSK3739937 SD 30 mg/ GSK3739937 SD 160 mg/SD PBO | Part 2 - Once Daily (QD) PBO | Part 2 (Cohort 3) - GSK3739937 QD 25 mg | Part 2 (Cohort 4) - GSK3739937 QD 50 mg | Part 2 (Cohort 5) - GSK3739937 QD 100 mg | Part 2 - Once Weekly (QW) PBO | Part 2 (Cohort 6) - GSK3739937 QW 500 mg | Part 3 (Cohort 7) - GSK3739937 PiB Fed/ GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted | Part 3 (Cohort 7) - GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed | Part 3 (Cohort 7) - GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed/ GSK3739937 Tablet Fed
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 4 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 (Cohort 1) - Single Dose (SD) Placebo (PBO)/GSK3739937 SD 80 mg/GSK3739937 SD 320 mg | Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ SD PBO/ GSK3739937 SD 320 mg | Part 1 (Cohort 1) - GSK3739937 SD 10 mg/ GSK3739937 SD 80 mg/SD PBO | Part 1 (Cohort 1) - GSK3739937 SD 800 mg | Part 1 (Cohort 1) - SD PBO | Part 1 (Cohort 2) - SD PBO/ GSK3739937 SD 160 mg/ GSK3739937 SD 640 mg | Part 1 (Cohort 2) - GSK3739937 SD 30mg/ SD PBO/ GSK3739937 SD 640mg | Part 1 (Cohort 2) - GSK3739937 SD 30 mg/ GSK3739937 SD 160 mg/SD PBO | Part 2 - Once Daily (QD) PBO | Part 2 (Cohort 3) - GSK3739937 QD 25 mg | Part 2 (Cohort 4) - GSK3739937 QD 50 mg | Part 2 (Cohort 5) - GSK3739937 QD 100 mg | Part 2 - Once Weekly (QW) PBO | Part 2 (Cohort 6) - GSK3739937 QW 500 mg | Part 3 (Cohort 7) - GSK3739937 PiB Fed/ GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted | Part 3 (Cohort 7) - GSK3739937 Tablet Fed/ GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed | Part 3 (Cohort 7) - GSK3739937 Tablet Fasted/ GSK3739937 PiB Fed/ GSK3739937 Tablet Fed | Total
Number analyzed (Participants) | 6 | 3 | 4 | 6 | 3 | 5 | 4 | 3 | 9 | 7 | 7 | 7 | 3 | 7 | 5 | 6 | 6 | 91
Age, Customized [Count of Participants; unit: Participants]
  <=18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  19-64 | 6 | 3 | 4 | 6 | 3 | 5 | 4 | 3 | 9 | 7 | 7 | 7 | 3 | 7 | 5 | 6 | 6 | 91
  >=65 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4
  Male | 4 | 3 | 4 | 6 | 3 | 5 | 4 | 3 | 8 | 7 | 7 | 6 | 3 | 7 | 5 | 6 | 6 | 87
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Central/South Asian Heritage | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian - Japanese Heritage | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 3 | 2 | 2 | 5 | 2 | 4 | 1 | 2 | 6 | 2 | 4 | 3 | 2 | 4 | 2 | 5 | 5 | 54
  Mixed Race | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  White - White/Caucasian/European Heritage | 3 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 3 | 3 | 3 | 4 | 0 | 3 | 3 | 1 | 1 | 32

OUTCOME MEASURES:

1. Primary Outcome: Part 1 - Number of Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect and important medical events may jeopardize the participant or may require medical or surgical intervention/Standard of care (SOC) to prevent one of the other outcomes mentioned before.
Time Frame: Up to 27 weeks
Population: Safety Population included all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Events
Groups:
- Placebo (PBO) Single Dose: In Cohort 1 and 2 of Part 1, participants received single oral dose of Placebo.
- GSK3739937 Single Dose (SD) 10 mg: In Cohort 1 of Part 1, participants received single oral dose of 10 mg GSK3739937
- GSK3739937 SD 30 mg: In Cohort 2 of Part 1, participants received single oral dose of 30 mg GSK3739937
- GSK3739937 SD 80 mg: In Cohort 1 of Part 1, participants received single oral dose of 80 mg GSK3739937
- GSK3739937 SD 160 mg: In Cohort 2 of Part 1, participants received single oral dose of 160 mg GSK3739937
- GSK3739937 SD 320 mg: In Cohort 1 of Part 1, participants received single oral dose of 320 mg GSK3739937
- GSK3739937 SD 640 mg: In Cohort 2 of Part 1, participants received single oral dose of 640 mg GSK3739937
- GSK3739937 SD 800 mg: In Cohort 1 of Part 1, participants received single oral dose of 800 mg of GSK3739937
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 21 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Events
  AEs | 7 | 1 | 3 | 3 | 0 | 2 | 4 | 2
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part 2 - Number of Any AEs and SAEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; is a congenital anomaly/birth defect and important medical events may jeopardize the participant or may require medical or surgical intervention/SOC to prevent one of the other outcomes mentioned before.
Time Frame: Up to 5 weeks
Population: Safety Population
Measure: Number; unit: Events
Groups:
- PBO Once Daily (QD): Participants received once daily doses of placebo for 14 days.
- GSK3739937 QD 25 mg: In Cohort 3 of Part 2, participants received once-daily oral dose of 25 mg GSK3739937 for 14 days.
- GSK3739937 QD 50 mg: In Cohort 4 of Part 2, participants received once-daily oral dose of 50 mg GSK3739937 for 14 days.
- GSK3739937 QD 100 mg: In Cohort 5 of Part 2, participants received once-daily oral dose of 100 mg GSK3739937 for 18 days.
- PBO Once Weekly (QW): Participants received once weekly oral dose of Placebo for over 3 weeks.
- GSK3739937 QW 500 mg: In Cohort 6 of Part 2, participants received one dose per week of 500 mg GSK3739937 for over 3 weeks.
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 9 | 7 | 7 | 7 | 3 | 7
Events
  AEs | 3 | 0 | 2 | 5 | 0 | 4
  SAEs | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Part 3 - Number of Any AEs and SAEs
Description: as for outcome 2
Time Frame: Up to 16 weeks
Population: Safety Population
Measure: Number; unit: Events
Groups:
- GSK3739937 PiB Fed: In Cohort 7 of Part 3, participants received single oral dose of 100 mg of GSK3739937 PiB as an oral suspension under moderate fed conditions in each one of the three periods.
- GSK3739937 Tablet Fed: In Cohort 7 of Part 3, participants received single oral dose of 100 mg of GSK3739937 Tablet under moderate fed conditions in each one of the three periods.
- GSK3739937 Tablet Fasted: In Cohort 7 of Part 3, participants received single oral dose of 100 mg of GSK3739937 Tablet under fasted conditions in each one of the three periods.
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
Events
  AEs | 2 | 4 | 6
  SAEs | 0 | 0 | 0

4. Primary Outcome: Part 1 - Change From Baseline in Hematology Parameters - Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets
Description: Blood samples were collected to assess change from baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelets. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9 cells/L)
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 18 | 1 | 6 | 6 | 6 | 6 | 6 | 6
Giga cells per liter (10^9 cells/L)
  Basophils | -0.01 (0.024) | 0 | 0 (0) | 0 (0) | -0.02 (0.041) | 0 (0) | 0 (0) | 0 (0)
  Eosinophils | -0.05 (0.092) | -0.2 | 0.02 (0.147) | -0.08 (0.075) | -0.02 (0.075) | -0.02 (0.041) | 0.08 (0.223) | -0.07 (0.082)
  Lymphocytes | 0.14 (0.391) | -0.5 | 0 (0.482) | -0.02 (0.248) | -0.13 (0.463) | 0.23 (0.339) | 0.25 (0.084) | -0.22 (0.248)
  Monocytes | 0.04 (0.124) | -0.1 | 0 (0.063) | -0.02 (0.194) | -0.03 (0.121) | 0.02 (0.133) | 0 (0.11) | -0.08 (0.117)
  Neutrophils | 0.3 (0.486) | 0.7 | 0.22 (0.306) | 0.08 (1.303) | 0.03 (0.468) | 0.33 (0.48) | 0.22 (0.117) | -0.03 (0.7)
  Platelets | 0.3 (26.73) | 2 | 8.2 (25.59) | 16 (27.71) | -6.3 (7.87) | 8.8 (20.5) | 13.2 (19.05) | 0.2 (13)

5. Primary Outcome: Part 2 (QD PBO and Cohort 3, 4 and 5) - Change From Baseline in Hematology Parameters - Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets
Description: as for outcome 4
Time Frame: Baseline (Day 1, pre-dose) and Day 14
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 9 | 7 | 3 | 6
10^9 cells/L
  Basophils | 0 (0) | 0 (0) | 0.03 (0.049) | -0.02 (0.041)
  Eosinophils | 0.03 (0.05) | -0.03 (0.095) | -0.01 (0.090) | 0.02 (0.075)
  Lymphocytes | -0.13 (0.26) | -0.07 (0.281) | 0.03 (0.427) | 0.15 (0.274)
  Monocytes | 0.02 (0.139) | 0.04 (0.113) | 0.01 (0.135) | -0.02 (0.117)
  Neutrophils | -0.47 (0.784) | -0.19 (0.682) | 0.03 (0.496) | -0.18 (0.877)
  Platelets | -11.9 (16.24) | -3.4 (18.12) | -9.7 (20.11) | -15.5 (32.93)

6. Primary Outcome: Part 2 (QW PBO and Cohort 6) - Change From Baseline in Hematology Parameters - Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets
Description: as for outcome 4
Time Frame: Baseline (Day 1, pre-dose) and Day 15
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 3 | 7
10^9 cells/L
  Basophils | 0 (0) | 0 (0)
  Eosinophils | 0.03 (0.115) | -0.01 (0.069)
  Lymphocytes | 0.23 (0.115) | 0.04 (0.378)
  Monocytes | 0.07 (0.058) | 0.06 (0.079)
  Neutrophils | -0.10 (0.173) | -0.27 (0.315)
  Platelets | -21.3 (47.72) | -9.3 (30.8)

7. Primary Outcome: Part 3 - Change From Baseline in Hematology Parameters - Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets
Description: as for outcome 4
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
10^9 cells/L
  Basophils | 0.01 (0.026) | 0 (0) | 0 (0)
  Eosinophils | -0.05 (0.052) | -0.05 (0.087) | -0.05 (0.092)
  Lymphocytes | 0.11 (0.253) | -0.08 (0.407) | 0.16 (0.184)
  Monocytes | 0.01 (0.099) | -0.01 (0.132) | 0.04 (0.083)
  Neutrophils | 0.16 (0.703) | -0.15 (1.253) | 0.17 (0.594)
  Platelets | 7 (15.83) | 1.5 (22.48) | -6.7 (21.4)

8. Primary Outcome: Part 1 - Change From Baseline in Hematology Parameters - Erythrocytes Count
Description: Blood samples were collected to assess change from baseline in Erythrocytes count. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Trillion cells per liter (10^12 cells/L)
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 18 | 1 | 6 | 6 | 6 | 6 | 6 | 6
Trillion cells per liter (10^12 cells/L) | 0.079 (0.1441) | 0.17 | 0.197 (0.3088) | 0.245 (0.1623) | 0.048 (0.2548) | 0.11 (0.1368) | 0.157 (0.1833) | 0.182 (0.1526)

9. Primary Outcome: Part 2 (QD PBO and Cohort 3, 4 and 5) - Change From Baseline in Hematology Parameters - Erythrocytes Count
Description: as for outcome 8
Time Frame: Baseline (Day 1, pre-dose) and Day 14
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 9 | 7 | 7 | 6
10^12 cells/L | -0.06 (0.1592) | 0.017 (0.175) | -0.227 (0.2423) | 0.037 (0.2601)

10. Primary Outcome: Part 2 (QW PBO and Cohort 6) - Change From Baseline in Hematology Parameters - Erythrocytes Count
Description: as for outcome 8
Time Frame: Baseline (Day 1, pre-dose) and Day 15
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 3 | 7
10^12 cells/L | -0.060 (0.2787) | -0.014 (0.1021)

11. Primary Outcome: Part 3 - Change From Baseline in Hematology Parameters - Erythrocytes Count
Description: as for outcome 8
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
10^12 cells/L | 0.229 (0.2193) | 0.197 (0.2287) | 0.189 (0.2014)

12. Primary Outcome: Part 1 - Change From Baseline in Hematology Parameter - Erythrocytes Mean Corpuscular Hemoglobin (MCH)
Description: Blood samples were collected to assess change from baseline in Erythrocytes Mean Corpuscular Hemoglobin (MCH). Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Picogram (pg)
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 18 | 1 | 6 | 6 | 6 | 6 | 6 | 6
Picogram (pg) | 0.09 (0.314) | -0.5 | 0.33 (0.294) | -0.08 (0.387) | -0.13 (0.32) | -0.13 (0.528) | -0.02 (0.232) | -0.03 (0.103)

13. Primary Outcome: Part 2 (QD PBO and Cohort 3, 4 and 5) - Change From Baseline in Hematology Parameter - Erythrocytes Mean Corpuscular Hemoglobin (MCH)
Description: as for outcome 12
Time Frame: Baseline (Day 1, pre-dose) and Day 14
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Picogram (pg)
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 9 | 7 | 7 | 6
Picogram (pg) | 0.02 (0.63) | -0.3 (0.44) | 0.16 (0.172) | -0.08 (0.605)

14. Primary Outcome: Part 2 (QW PBO and Cohort 6) - Change From Baseline in Hematology Parameter - Erythrocytes Mean Corpuscular Hemoglobin (MCH)
Description: Blood samples were collected to assess change from baseline in Mean Corpuscular Hemoglobin (MCH). Blood samples were collected to assess change from baseline in Erythrocytes Mean Corpuscular Hemoglobin (MCH). Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, pre-dose) and Day 15
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Picogram (pg)
Arm/Group | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 3 | 7
Picogram (pg) | -0.87 (0.666) | -0.83 (0.399)

15. Primary Outcome: Part 3 - Change From Baseline in Hematology Parameter - Erythrocytes Mean Corpuscular Hemoglobin (MCH)
Description: as for outcome 14
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Picogram (pg)
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
Picogram (pg) | 0 (0.433) | -0.24 (0.487) | 0.05 (0.54)

16. Primary Outcome: Part 1 - Change From Baseline in Hematology Parameter - Hematocrit
Description: Blood samples were collected to assess change from baseline in Hematocrit. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 18 | 1 | 6 | 6 | 6 | 6 | 6 | 6
Proportion of red blood cells in blood | 0.0083 (0.01231) | 0.014 | 0.015 (0.0304) | 0.0237 (0.01491) | 0.0012 (0.02409) | 0.0047 (0.00866) | 0.0117 (0.01862) | 0.0175 (0.01319)

17. Primary Outcome: Part 2 (QD PBO and Cohort 3, 4 and 5) - Change From Baseline in Hematology Parameter - Hematocrit
Description: as for outcome 16
Time Frame: Baseline (Day 1, pre-dose) and Day 14
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 9 | 7 | 7 | 6
Proportion of red blood cells in blood | -0.0081 (0.01342) | 0.0066 (0.01838) | -0.0217 (0.01963) | 0.0043 (0.01929)

18. Primary Outcome: Part 2 (QW PBO and Cohort 6) - Change From Baseline in Hematology Parameter - Hematocrit
Description: as for outcome 16
Time Frame: Baseline (Day 1, pre-dose) and Day 15
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 3 | 7
Proportion of red blood cells in blood | -0.0120 (0.02685) | -0.0094 (0.00781)

19. Primary Outcome: Part 3 - Change From Baseline in Hematology Parameter - Hematocrit
Description: as for outcome 16
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
Proportion of red blood cells in blood | 0.0182 (0.01826) | 0.013 (0.02076) | 0.0159 (0.01793)

20. Primary Outcome: Part 1 - Change From Baseline in Hematology Parameter - Reticulocytes
Description: Blood samples were collected to assess change from baseline in Reticulocytes. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of reticulocytes in blood
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 18 | 1 | 6 | 6 | 6 | 6 | 6 | 6
Proportion of reticulocytes in blood | 0.0008 (0.00363) | 0.002 | -0.0045 (0.00622) | -0.0008 (0.00264) | -0.0007 (0.00234) | -0.0015 (0.00302) | -0.0008 (0.00194) | -0.0008 (0.0016)

21. Primary Outcome: Part 2 (QD PBO and Cohort 3, 4 and 5) - Change From Baseline in Hematology Parameter - Reticulocytes
Description: as for outcome 20
Time Frame: Baseline (Day 1, pre-dose) and Day 14
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of reticulocytes in blood
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 9 | 7 | 7 | 6
Proportion of reticulocytes in blood | -0.0017 (0.0024) | -0.0011 (0.00219) | 0.0010 (0.00306) | -0.0012 (0.00264)

22. Primary Outcome: Part 2 (QW PBO and Cohort 6) - Change From Baseline in Hematology Parameter - Reticulocytes
Description: as for outcome 20
Time Frame: Baseline (Day 1, pre-dose) and Day 15
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of reticulocytes in blood
Arm/Group | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 3 | 7
Proportion of reticulocytes in blood | 0.0003 (0.00379) | -0.0001 (0.00227)

23. Primary Outcome: Part 3 - Change From Baseline in Hematology Parameter - Reticulocytes
Description: as for outcome 20
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Proportion of reticulocytes in blood
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
Proportion of reticulocytes in blood | -0.0011 (0.00231) | -0.0009 (0.00255) | -0.0012 (0.00224)

24. Primary Outcome: Part 1 - Change From Baseline in Hematology Parameter - Hemoglobin (Hb)
Description: Blood samples were collected to assess change from baseline in Hemoglobin (Hb). Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 18 | 1 | 6 | 6 | 6 | 6 | 6 | 6
Grams per liter (g/L) | 2.8 (4.44) | 2 | 7.5 (8.41) | 6.7 (5.2) | 1 (8.51) | 2.7 (2.73) | 4.3 (5.68) | 5.2 (4.07)

25. Primary Outcome: Part 2 (QD PBO and Cohort 3, 4 and 5) - Change From Baseline in Hematology Parameter - Hemoglobin (Hb)
Description: as for outcome 24
Time Frame: Baseline (Day 1, pre-dose) and Day 14
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 9 | 7 | 7 | 6
Grams per liter (g/L) | -1.6 (5.13) | -1 (7.21) | -5.7 (6.70) | 0.5 (7.74)

26. Primary Outcome: Part 2 (QW PBO and Cohort 6) - Change From Baseline in Hematology Parameter - Hemoglobin (Hb)
Description: as for outcome 24
Time Frame: Baseline (Day 1, pre-dose) and Day 15
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 3 | 7
Grams per liter (g/L) | -5.7 (7.64) | -4.3 (2.63)

27. Primary Outcome: Part 3 - Change From Baseline in Hematology Parameter - Hemoglobin (Hb)
Description: as for outcome 24
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
Grams per liter (g/L) | 6.7 (5.87) | 4.5 (7.07) | 5.7 (5.37)

28. Primary Outcome: Part 1 - Change From Baseline in Clinical Chemistry Parameter - Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphate (ALP) and Serum Creatine Phosphokinase (CPK)
Description: Blood samples were collected to assess change from baseline in Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphate (ALP) and Serum Creatine Phosphokinase (CPK). Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter (IU/L)
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 18 | 1 | 6 | 6 | 6 | 6 | 6 | 6
International units per Liter (IU/L)
  ALP | 4.6 (6.06) | 5 | 8.3 (4.27) | 6.7 (3.72) | 3 (3.95) | 6.2 (4.92) | 8.8 (8.04) | 6.2 (2.14)
  ALT | 1.6 (7.78) | -1 | -4.2 (6.05) | -0.8 (3.49) | 0.3 (9.35) | -3.5 (6.32) | 1.2 (10.19) | -1.3 (3.39)
  AST | -1.5 (6.07) | -8 | -4.5 (4.93) | -2 (2.83) | -0.5 (4.04) | -3.8 (4.26) | -1.8 (4.79) | -1.5 (3.02)
  CPK: number analyzed (Participants) | 6 | 1 | 6 | 6 | 6 | 6 | 4 | 6
  CPK | -29.3 (140.65) | 0.776 | -0.1978 (0.48809) | -0.0777 (0.72185) | -0.1292 (0.91507) | 0.2242 (0.3425) | -60.5 (132.53) | -20 (39.47)

29. Primary Outcome: Part 2 (QD PBO and Cohort 3, 4 and 5) - Change From Baseline in Clinical Chemistry Parameter - ALT, AST, ALP and Serum CPK
Description: as for outcome 28
Time Frame: Baseline (Day 1, pre-dose) and Day 14
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter (IU/L)
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 9 | 7 | 7 | 6
International units per Liter (IU/L)
  ALP | -0.4 (14.44) | -4.6 (10.61) | 5.9 (5.34) | 3.0 (9.76)
  ALT | -3.1 (6.9) | -5.9 (5.84) | -3.9 (7.10) | 0.3 (4.27)
  AST | -4.6 (5.2) | -7.1 (5.52) | -4.1 (4.53) | 3.2 (3.25)
  CPK: number analyzed (Participants) | 6 | 0 | 7 | 6
  CPK | -1 (26.43) |  | 19.4 (88.50) | 14.8 (41.63)

30. Primary Outcome: Part 2 (QW PBO and Cohort 6) - Change From Baseline in Clinical Chemistry Parameter -ALT, AST, ALP and Serum CPK
Description: as for outcome 28
Time Frame: Baseline (Day 1, pre-dose) and Day 15
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter (IU/L)
Arm/Group | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 3 | 7
International units per Liter (IU/L)
  ALP | 0.0 (2.65) | 1.9 (4.02)
  ALT | -2.3 (7.77) | -3.1 (2.91)
  AST | -3.0 (2.65) | -3 (1.83)
  CPK | -18.7 (14.84) | -22.6 (35.72)

31. Primary Outcome: Part 3 - Change From Baseline in Clinical Chemistry Parameter - ALT, AST, ALP and CPK
Description: as for outcome 28
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: International units per Liter (IU/L)
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
International units per Liter (IU/L)
  ALP | 5.9 (6.42) | 5.4 (5.91) | 5.2 (4.78)
  ALT | 1.3 (4.32) | -0.2 (4.92) | -0.4 (3.16)
  AST | 0.3 (3.67) | 0.4 (4.4) | -0.9 (3.02)
  CPK | -27.3 (52.49) | -22.2 (45.6) | -62.1 (73.59)

32. Primary Outcome: Part 1 - Change From Baseline in Clinical Chemistry Parameters- Bicarbonate, Calcium, Glucose, Chloride, Magnesium, Phosphate, Potassium, Sodium, Blood Urea Nitrogen, Cholesterol, High Density Lipoprotein, Low Density Lipoprotein, Triglycerides
Description: Blood samples were collected to assess change from baseline in Bicarbonate, Calcium, Glucose, Chloride, Magnesium, Phosphate, Potassium, Sodium, Blood Urea Nitrogen (BUN), Cholesterol, High Density Lipoprotein (HDL), Low Density Lipoprotein (LDL) and Triglycerides. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (mmol/L)
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 18 | 1 | 6 | 6 | 6 | 6 | 6 | 6
Millimoles per Liter (mmol/L)
  Glucose | -0.29 (0.46027) | -0.499 | -0.3147 (0.22689) | -0.1387 (0.36972) | -0.157 (0.22077) | -0.379 (0.22041) | -0.1848 (0.25449) | -0.3147 (0.25488)
  Bicarbonate | 1.8 (2.62) | 2 | 1.8 (2.48) | 3.3 (3.5) | 1.7 (1.97) | -0.2 (2.14) | 0.7 (2.25) | 1.3 (1.51)
  Calcium | 0.0693 (0.10417) | -0.025 | 0.0208 (0.10249) | 0.1453 (0.04816) | 0.0707 (0.13915) | 0.0208 (0.10888) | 0.2203 (0.17728) | 0.0375 (0.05646)
  Cholesterol | 0.1294 (0.59228) | 0.104 | -0.2627 (0.52795) | 0.444 (0.16643) | -0.224 (0.87169) | 0.0047 (0.5061) | 0.1898 (0.3552) | 0.142 (0.09784)
  Chloride | -1.6 (2.79) | -1 | -0.3 (1.75) | -5 (1.41) | 1.7 (1.51) | -1.3 (1.51) | -0.8 (1.83) | 0.3 (1.03)
  HDL | -0.0187 (0.20182) | 0.181 | -0.069 (0.20186) | 0.1247 (0.15293) | -0.086 (0.13432) | 0.082 (0.11534) | -0.0388 (0.30208) | -0.043 (0.07956)
  Potassium | -0.02 (0.303) | -0.2 | 0.18 (0.354) | 0.18 (0.293) | 0.1 (0.261) | -0.28 (0.24) | -0.07 (0.234) | -0.12 (0.214)
  LDL | -0.0027 (0.44009) | -0.078 | -0.0605 (0.51701) | 0.5217 (0.21608) | -0.5298 (0.52526) | 0.004 (0.35306) | 0.2023 (0.22274) | -0.0388 (0.29351)
  Magnesium | 0.0046 (0.05426) | 0 | -0.0137 (0.06173) | 0.0068 (0.03086) | -0.0478 (0.03086) | 0.0752 (0.06035) | 0.0342 (0.03086) | 0.0137 (0.02117)
  Phosphate | 0.0611 (0.13184) | 0.097 | 0.0377 (0.1266) | 0.124 (0.13169) | -0.0108 (0.16164) | 0.0052 (0.08782) | 0.043 (0.12387) | -0.0108 (0.05669)
  Sodium | 0 (1.64) | 0 | 1 (1.26) | 0.2 (0.98) | 1 (1.26) | -0.7 (1.51) | -0.3 (1.37) | 2.2 (0.98)
  Triglycerides | 0.1683 (0.46481) | 0.18 | -0.2225 (0.43845) | 0.0318 (0.41469) | -0.2337 (0.3573) | -0.0863 (0.32709) | 0.087 (0.12521) | 0.1467 (0.25766)
  BUN | -0.2777 (0.7798) | 1.071 | -0.4165 (0.79561) | 0.2975 (0.7629) | -0.119 (0.62517) | 0.2975 (0.47451) | -0.2975 (0.72872) | -0.595 (0.29149)

33. Primary Outcome: Part 2 (QD PBO and Cohort 3, 4 and 5) - Change From Baseline in Clinical Chemistry Parameters- Bicarbonate, Calcium, Glucose, Chloride, Magnesium, Phosphate, Potassium, Sodium, BUN, Cholesterol, HDL, LDL, Triglycerides
Description: as for outcome 32
Time Frame: Baseline (Day 1, pre-dose) and Day 14
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (mmol/L)
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 9 | 7 | 7 | 6
Millimoles per Liter (mmol/L)
  Glucose | -0.2773 (0.58989) | -0.6027 (0.19341) | 0.0319 (0.35520) | -0.3978 (0.24715)
  Bicarbonate | -1 (1.94) | -1.4 (1.4) | -0.6 (2.44) | -0.3 (2.07)
  Calcium | -0.0306 (0.14997) | -0.2136 (0.12771) | -0.0286 (0.08469) | 0.0373 (0.07016)
  Cholesterol | -0.2701 (0.56002) | -0.6503 (0.68612) | -0.2843 (0.42535) | 0.3708 (0.43447)
  Chloride | 0.3 (2.5) | 3 (1.15) | -1.0 (1.63) | -1.3 (2.16)
  HDL | -0.1438 (0.15951) | -0.1849 (0.13459) | -0.0777 (0.14711) | -0.0948 (0.21847)
  Potassium | -0.09 (0.44) | -0.29 (0.261) | 0 (0.191) | -0.22 (0.449)
  LDL | -0.2902 (0.38135) | -0.5244 (0.48959) | -0.2807 (0.30973) | -0.0903 (0.86478)
  Magnesium | -0.0547 (0.09168) | -0.0996 (0.06635) | -0.0527 (0.05659) | -0.0205 (0.06737)
  Phosphate | -0.0573 (0.12367) | -0.1477 (0.10973) | 0.0831 (0.11469) | 0.0485 (0.09964)
  Sodium | 0.6 (1.67) | 1.3 (0.76) | -0.9 (1.07) | 0.3 (1.97)
  Triglycerides | 0.0403 (0.20877) | -0.1614 (0.26907) | 0.0434 (0.20744) | 0.2577 (0.33429)
  BUN | 0.0397 (0.9849) | 0.408 (0.90851) | -0.1020 (1.02466) | 0.1190 (0.53748)

34. Primary Outcome: Part 2 (QW PBO and Cohort 6) - Change From Baseline in Clinical Chemistry Parameters- Bicarbonate, Calcium, Glucose, Chloride, Magnesium, Phosphate, Potassium, Sodium, BUN, Cholesterol, HDL, LDL, Triglycerides
Description: as for outcome 32
Time Frame: Baseline (Day 1, pre-dose) and Day 15
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (mmol/L)
Arm/Group | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 3 | 7
Millimoles per Liter (mmol/L)
  Glucose | -0.2590 (0.23106) | -0.3014 (0.14978)
  Bicarbonate | -0.7 (2.08) | -0.3 (1.38)
  Calcium | -0.0913 (0.14160) | -0.0391 (0.10029)
  Cholesterol | -0.4483 (0.39167) | -0.203 (0.56917)
  Chloride | 1.3 (0.58) | 0.4 (1.62)
  HDL | -0.1037 (0.11860) | -0.0703 (0.14776)
  Potassium | -0.10 (0.346) | -0.21 (0.418)
  LDL | -0.4137 (0.34187) | -0.1107 (0.36147)
  Magnesium | 0.0137 (0.02367) | 0.0059 (0.04981)
  Phosphate | 0.0540 (0.10437) | 0.0464 (0.08088)
  Sodium | -0.3 (1.15) | -0.7 (1.5)
  Triglycerides | 0.0267 (0.07243) | 0.0129 (0.25175)
  BUN | 0.1190 (0.54533) | 0.408 (0.32121)

35. Primary Outcome: Part 3 - Change From Baseline in Clinical Chemistry Parameters- Bicarbonate, Calcium, Glucose, Chloride, Magnesium, Phosphate, Potassium, Sodium, BUN, Cholesterol, HDL, LDL, Triglycerides Edit Properties | Duplicate Measure
Description: as for outcome 32
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per Liter (mmol/L)
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
Millimoles per Liter (mmol/L)
  Glucose | -0.2033 (0.39) | -0.3755 (0.24961) | -0.2145 (0.27017)
  Bicarbonate | 1.5 (1.96) | 0.4 (2.12) | 1.5 (1.64)
  Calcium | 0.055 (0.10971) | 0.0793 (0.10607) | 0.0666 (0.07293)
  Cholesterol | 0.1087 (0.30739) | 0.1218 (0.3317) | 0.0569 (0.47643)
  Chloride | -1.2 (2.57) | -2.2 (2.14) | -1.6 (1.92)
  HDL | -0.0259 (0.13992) | -0.0549 (0.12044) | -0.0415 (0.1084)
  Potassium | -0.03 (0.422) | -0.04 (0.361) | -0.17 (0.364)
  LDL | 0.219 (0.42617) | 0.2312 (0.46471) | 0.0484 (0.55487)
  Magnesium | 0.0109 (0.07972) | 0.0217 (0.06338) | 0.0109 (0.0883)
  Phosphate | -0.0021 (0.11269) | -0.0058 (0.07409) | -0.0021 (0.0965)
  Sodium | 0.5 (2.47) | -1.1 (1.45) | 0.3 (1.95)
  Triglycerides | 0.1558 (0.44508) | 0.1801 (0.37021) | 0.0082 (0.30805)
  BUN | 0.6426 (0.91715) | 0.504 (0.81856) | 0.4046 (1.00855)

36. Primary Outcome: Part 1 - Change From Baseline in Clinical Chemistry Parameters - Amylase and Lipase
Description: Blood samples were collected to assess change from baseline in Amylase and Lipase. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 18 | 1 | 6 | 6 | 6 | 6 | 6 | 6
Units per liter (U/L)
  Amylase | -1.2 (17.38) | 12 | -0.7 (6.12) | -0.7 (4.46) | 3.7 (4.76) | 5.8 (12.02) | -1.7 (11.52) | 3.7 (17.24)
  Lipase | 7.8 (25.41) | -31 | -15.5 (25.76) | -8 (20.01) | -1.3 (3.93) | 3.7 (3.67) | 3.7 (4.27) | 3.8 (5.19)

37. Primary Outcome: Part 2 (QD PBO and Cohort 3, 4 and 5) - Change From Baseline in Clinical Chemistry Parameters - Amylase and Lipase
Description: as for outcome 36
Time Frame: Baseline (Day 1, pre-dose) and Day 14
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 9 | 7 | 7 | 6
Units per liter (U/L)
  Amylase | 3.7 (27.96) | -18.3 (17.85) | 0.3 (5.50) | 7.2 (15.30)
  Lipase | 3.8 (22.06) | -6.3 (8.62) | 1.1 (2.54) | 1.2 (2.48)

38. Primary Outcome: Part 2 (QW PBO and Cohort 6) - Change From Baseline in Clinical Chemistry Parameters - Amylase and Lipase
Description: as for outcome 36
Time Frame: Baseline (Day 1, pre-dose) and Day 15
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 3 | 7
Units per liter (U/L)
  Amylase | 2.7 (7.51) | -10 (22.5)
  Lipase | -2.0 (5.57) | -1.9 (4.67)

39. Primary Outcome: Part 3 - Change From Baseline in Clinical Chemistry Parameters - Amylase and Lipase
Description: as for outcome 36
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
Units per liter (U/L)
  Amylase | 0.5 (16.41) | 1.2 (12.08) | 5.1 (18.24)
  Lipase | 0.4 (18.92) | -0.6 (6.25) | 2.7 (10.06)

40. Primary Outcome: Part 1 - Change From Baseline in Clinical Chemistry Parameter - Total Bilirubin, Direct Bilirubin and Creatinine
Description: Blood samples were collected to assess change from baseline in Total Bilirubin, Direct Bilirubin and Creatinine. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per Liter (umol/L)
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 18 | 1 | 6 | 6 | 6 | 6 | 6 | 6
Micromoles per Liter (umol/L)
  Direct Bilirubin | -0.2839 (1.10348) | 0 | -0.1995 (0.62518) | 0.4895 (0.46819) | -0.285 (1.28724) | 0.2565 (1.18349) | -0.3705 (0.86801) | -0.855 (1.43069)
  Total Bilirubin | -0.19 (3.2598) | -1.71 | -0.855 (2.8098) | 0.57 (0.883) | 0.285 (2.5171) | 0.285 (2.7396) | -1.71 (2.163) | -3.135 (3.8109)
  Creatinine | 1.8171 (5.38547) | -8.84 | 6.188 (8.27379) | 6.0407 (3.93024) | 4.5673 (8.82968) | -0.442 (3.65553) | 3.978 (4.80135) | 3.536 (2.56208)

41. Primary Outcome: Part 2 (QD PBO and Cohort 3, 4 and 5) - Change From Baseline in Clinical Chemistry Parameter - Total Bilirubin, Direct Bilirubin and Creatinine
Description: as for outcome 40
Time Frame: Baseline (Day 1, pre-dose) and Day 14
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per Liter (umol/L)
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 9 | 7 | 7 | 6
Micromoles per Liter (umol/L)
  Direct Bilirubin | -0.6058 (1.12324) | 0.5863 (1.10758) | -0.8061 (0.95062) | 0.2817 (1.28814)
  Total Bilirubin | 0.19 (3.9593) | 0.244 (3.6178) | -0.977 (2.7674) | 1.425 (3.8109)
  Creatinine | 3.536 (7.48795) | -1.768 (5.35289) | -0.6314 (4.55680) | 8.3980 (2.89164)

42. Primary Outcome: Part 2 (QW PBO and Cohort 6) - Change From Baseline in Clinical Chemistry Parameter - Total Bilirubin, Direct Bilirubin and Creatinine
Description: as for outcome 40
Time Frame: Baseline (Day 1, pre-dose) and Day 15
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per Liter (umol/L)
Arm/Group | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 3 | 7
Micromoles per Liter (umol/L)
  Direct Bilirubin | 0.5700 (0.98727) | 1.4671 (0.64254)
  Total Bilirubin | -1.140 (2.6121) | 1.71 (1.71)
  Creatinine | -1.1787 (2.55189) | 2.2731 (2.88068)

43. Primary Outcome: Part 3 - Change From Baseline in Clinical Chemistry Parameter - Total Bilirubin, Direct Bilirubin and Creatinine
Description: as for outcome 40
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per Liter (umol/L)
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
Micromoles per Liter (umol/L)
  Direct Bilirubin | 0.3306 (0.89198) | 0.4124 (1.068) | 0.2059 (1.11784)
  Total Bilirubin | 0.456 (1.9886) | 0.905 (3.7813) | 1.026 (3.5282)
  Creatinine | 3.0645 (6.90318) | 1.716 (6.168) | 2.9467 (6.70465)

44. Primary Outcome: Part 1 - Change From Baseline in Clinical Chemistry Parameter - Total Protein
Description: Blood samples were collected to assess change from baseline in Total Protein. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Grams per Liter (g/L)
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 18 | 1 | 6 | 6 | 6 | 6 | 6 | 6
Grams per Liter (g/L) | 3.2 (3.07) | 2 | 4.5 (3.83) | 6.3 (3.33) | 1 (4.15) | 3.7 (2.88) | 4 (3.85) | 3.5 (1.97)

45. Primary Outcome: Part 2 - (QD PBO and Cohort 3, 4 and 5) - Change From Baseline in Clinical Chemistry Parameter - Total Protein
Description: as for outcome 44
Time Frame: Baseline (Day 1, pre-dose) and Day 14
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Grams per Liter (g/L)
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 9 | 7 | 7 | 6
Grams per Liter (g/L) | -3.7 (3.84) | -7.1 (6.26) | -5.4 (3.91) | 2.0 (2.83)

46. Primary Outcome: Part 2 (QW PBO and Cohort 6) - Change From Baseline in Clinical Chemistry Parameter - Total Protein
Description: as for outcome 44
Time Frame: Baseline (Day 1, pre-dose) and Day 15
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Grams per Liter (g/L)
Arm/Group | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 3 | 7
Grams per Liter (g/L) | -1.7 (5.03) | -2.1 (4.49)

47. Primary Outcome: Part 3 - Change From Baseline in Clinical Chemistry Parameter - Total Protein
Description: as for outcome 44
Time Frame: Baseline (Day -1) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Grams per Liter (g/L)
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
Grams per Liter (g/L) | 5.1 (5.38) | 5.4 (4.87) | 4.5 (4.02)

48. Primary Outcome: Part 1 - Number of Participants With Abnormal Urinalysis Parameters
Description: Urine samples were collected to detect presence of occult blood and protein through dipstick and random method respectively. The results presented are worst case abnormal urinalysis results post-baseline relative to baseline.
Time Frame: Up to 27 weeks
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 21 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Occult Blood | 4 | 0 | 1 | 1 | 2 | 3 | 1 | 2
  Protein | 2 | 2 | 2 | 1 | 0 | 1 | 0 | 1

49. Primary Outcome: Part 2 - Number of Participants With Abnormal Urinalysis Parameters
Description: as for outcome 48
Time Frame: Up to 5 weeks
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 9 | 7 | 7 | 7 | 3 | 7
Participants
  Occult Blood | 2 | 1 | 3 | 0 | 1 | 3
  Protein | 1 | 0 | 2 | 0 | 1 | 1

50. Primary Outcome: Part 3 - Number of Participants With Abnormal Urinalysis Parameters
Description: as for outcome 48
Time Frame: Up to 16 weeks
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
Participants
  Occult Blood | 1 | 1 | 1
  Protein | 4 | 2 | 2

51. Primary Outcome: Part 1 - Change From Baseline in Vital Signs: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: Blood pressure (SBP and DBP) was assessed in semi-supine position with a completely automated device. Blood pressure measurement preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline is defined as the average of the triplicate predose assessments within each treatment. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, pre-dose) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 18 | 1 | 6 | 6 | 6 | 6 | 6 | 6
Millimeters of mercury (mmHg)
  SBP | 5.3 (7.82) | 0.5 | -0.1 (14.68) | 4.6 (7.07) | 2.3 (7.30) | 1.3 (8.04) | 2.4 (6.34) | 5.5 (8.95)
  DBP | 4.0 (4.36) | 1.8 | 3.0 (8.20) | 3.7 (9.57) | 1.7 (6.15) | -1.2 (4.05) | 2.7 (8.13) | 4.7 (7.06)

52. Primary Outcome: Part 2 (QD PBO and Cohort 3, 4 and 5) - Change From Baseline in Vital Signs - Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: as for outcome 51
Time Frame: Baseline (Day 1, pre-dose) and Day 14
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 9 | 7 | 7 | 7
Millimeters of mercury (mmHg)
  SBP | -6.0 (15.26) | -2.1 (11.58) | -2.1 (5.57) | -0.8 (4.08)
  DBP | -3.4 (8.73) | 0.8 (7.21) | 1.4 (5.45) | 0.0 (6.17)

53. Primary Outcome: Part 2 (QW PBO and Cohort 6) - Change From Baseline in Vital Signs - Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: as for outcome 51
Time Frame: Baseline (Day 1, pre-dose) and Day 15
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 3 | 7
Millimeters of mercury (mmHg)
  SBP | 1.0 (11.89) | 1.5 (5.42)
  DBP | 4.2 (9.56) | 0.9 (6.52)

54. Primary Outcome: Part 3 - Change From Baseline in Vital Signs - Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: as for outcome 51
Time Frame: Baseline (Day 1, pre-dose) and Day 6
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
Millimeters of mercury (mmHg)
  SBP | 6.2 (7.20) | 3.8 (10.10) | 9.3 (8.08)
  DBP | 2.3 (4.02) | 3.4 (8.63) | 4.4 (5.79)

55. Primary Outcome: Part 1 - Change From Baseline in Vital Signs - Pulse Rate
Description: Pulse rate was assessed in semi-supine position with a completely automated device. Pulse rate measurement preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, pre-dose) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 18 | 1 | 6 | 6 | 6 | 6 | 6 | 6
Beats per minute | 1.5 (5.03) | 15.7 | 3.5 (7.40) | -0.2 (3.45) | 5.9 (2.64) | 4.8 (5.74) | -0.9 (7.98) | 0.0 (9.71)

56. Primary Outcome: Part 2 (QD PBO and Cohort 3, 4 and 5) - Change From Baseline in Vital Signs - Pulse Rate
Description: as for outcome 55
Time Frame: Baseline (Day 1, pre-dose) and Day 14
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 9 | 7 | 7 | 6
Beats per minute | 1.1 (4.59) | -2.8 (4.98) | 5.0 (5.49) | 3.0 (4.75)

57. Primary Outcome: Part 2 (QW PBO and Cohort 6) - Change From Baseline in Vital Signs - Pulse Rate
Description: as for outcome 55
Time Frame: Baseline (Day 1, pre-dose) and Day 15
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 3 | 7
Beats per minute | 0.9 (1.60) | 5.2 (5.29)

58. Primary Outcome: Part 3 - Change From Baseline in Vital Signs - Pulse Rate
Description: as for outcome 55
Time Frame: Baseline (Day 1, pre-dose) and Day 6
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
Beats per minute | 6.2 (6.80) | 7.4 (4.98) | 6.6 (5.48)

59. Primary Outcome: Part 1 - Change From Baseline in Vital Signs - Body Temperature
Description: Temperature was assessed in the semi-recumbent position with a completely automated device, preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, pre-dose) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 18 | 1 | 6 | 6 | 6 | 6 | 6 | 6
Degrees Celsius | -0.06 (0.320) | -0.10 | 0.12 (0.248) | -0.05 (0.226) | 0.10 (0.190) | 0.02 (0.117) | 0.08 (0.286) | 0.20 (0.155)

60. Primary Outcome: Part 2 (QD PBO and Cohort 3, 4 and 5) - Change From Baseline in Vital Signs - Body Temperature
Description: Body temperature were assessed at indicated time-points. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, pre-dose) and Day 14
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 9 | 7 | 7 | 7
Degrees Celsius | 0.16 (0.283) | -0.07 (0.170) | 0.09 (0.135) | -0.08 (0.204)

61. Primary Outcome: Part 2 (QW PBO and Cohort 6) - Change From Baseline in Vital Signs - Body Temperature
Description: as for outcome 60
Time Frame: Baseline (Day 1, pre-dose) and Day 15
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 3 | 7
Degrees Celsius | -0.07 (0.153) | -0.06 (0.113)

62. Primary Outcome: Part 3 - Change From Baseline in Vital Signs - Body Temperature
Description: as for outcome 60
Time Frame: Baseline (Day 1, pre-dose) and Day 6
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
Degrees Celsius | 0.08 (0.231) | 0.06 (0.237) | 0.15 (0.233)

63. Primary Outcome: Part 1 - Change From Baseline in Vital Signs - Respiratory Rate
Description: Respiratory rate was assessed in the semi-recumbent position with a completely automated device, preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline value is presented and was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, pre-dose) and Day 6
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 21 | 1 | 6 | 6 | 6 | 6 | 6 | 6
Breaths per minute | 0.7 (2.97) | -5.0 | -3.0 (1.41) | 3.7 (1.03) | 0.7 (2.07) | 0.3 (1.51) | 0.3 (1.51) | 0.7 (3.27)

64. Primary Outcome: Part 2 (QD PBO and Cohort 3, 4 and 5) - Change From Baseline in Vital Signs - Respiratory Rate
Description: as for outcome 63
Time Frame: Baseline (Day 1, pre-dose) and Day 14
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 9 | 7 | 7 | 7
Breaths per minute | -0.4 (2.19) | -3.4 (1.51) | 0.0 (1.63) | 1.2 (3.13)

65. Primary Outcome: Part 2 (QW PBO and Cohort 6) - Change From Baseline in Vital Signs - Respiratory Rate
Description: as for outcome 63
Time Frame: Baseline (Day 1, pre-dose) and Day 15
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 3 | 7
Breaths per minute | 0.0 (2.00) | -1.4 (2.23)

66. Primary Outcome: Part 3 - Change From Baseline in Vital Signs - Respiratory Rate
Description: as for outcome 63
Time Frame: Baseline (Day 1, pre-dose) and Day 6
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
Breaths per minute | 0.4 (2.03) | -0.3 (2.31) | 1.2 (2.24)

67. Primary Outcome: Part 1 - Number of Participants With Worst Case Post-Baseline Electrocardiogram (ECG) Findings
Description: Twelve lead ECGs were obtained using an ECG machine that automatically calculated the heart rate and measured PR, QRS, QT, and QT interval corrected using the Fridericia's formula (QTcF) intervals. ECG findings were categorized as Normal, Abnormal clinically significant (CS) and Abnormal not clinically significant (NCS). Clinically significant abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. Data for number of participants with worst case post-Baseline ECG findings have been presented.
Time Frame: Up to 27 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 21 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Participants
  Normal | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
  Abnormal - Not Clinically Significant | 20 | 4 | 6 | 6 | 6 | 5 | 6 | 6
  Abnormal - Clinically Significant | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

68. Primary Outcome: Part 2 - Number of Participants With Worst Case Post-Baseline ECG Findings
Description: as for outcome 67
Time Frame: Up to 5 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg | PBO Once Weekly (QW) | GSK3739937 QW 500 mg
Number analyzed (Participants) | 9 | 7 | 7 | 7 | 3 | 7
Participants
  Normal | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal - Not Clinically Significant | 9 | 7 | 7 | 7 | 3 | 7
  Abnormal - Clinically Significant | 0 | 0 | 0 | 0 | 0 | 0

69. Primary Outcome: Part 3 - Number of Participants With Worst Case Post-Baseline ECG Findings
Description: as for outcome 67
Time Frame: Up to 16 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 17 | 15
Participants
  Normal | 1 | 1 | 1
  Abnormal - Not Clinically Significant | 14 | 16 | 14
  Abnormal - Clinically Significant | 0 | 0 | 0

70. Primary Outcome: Part 3 - Area Under the Plasma Concentration Time Curve (AUC) From Zero to 24 Hours (AUC[0-24]) of GSK3739937
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of GSK3739937. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 12, 16 and 24 hours post-dose in each treatment period
Population: Pharmacokinetic (PK) Population: The PK Population included all participants who undergo plasma or urine PK sampling and have evaluable PK assay results. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanogram/ millilitre (h*ng/mL)
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 16 | 15
Hour*nanogram/ millilitre (h*ng/mL) | 6455.362 (25) | 8646.757 (33.9) | 3522.969 (91)
Statistical Analysis 1: Comparison: GSK3739937 Tablet Fed vs GSK3739937 Tablet Fasted; The mixed model was used to estimate Food Effect for the log transformed parameter AUC (0-24). Analysis was performed using fed/ fasted state and tablet/ PiB as fixed effects and participant as a random effect; Test type: Other; Mixed Models Analysis; Geometric Least Square Mean Ratio = 2.462, 90% CI 2-sided [1.823 to 3.323]
Statistical Analysis 2: Comparison: GSK3739937 PiB Fed vs GSK3739937 Tablet Fed; The mixed model was used to estimate Tablet vs. PiB effect for the log transformed parameter AUC (0-24). Analysis was performed using the independent variables included a fixed effect for treatment (PiB or Tablet) and period, and participant as a random effect; Test type: Other; Mixed Models Analysis; Geometric Least Square Mean Ratio = 1.381, 90% CI 2-sided [1.223 to 1.56]

71. Primary Outcome: Part 3 - AUC From Time Zero (Pre-dose) Extrapolated to Infinite Time (AUC[0-inf]) of GSK3739937
Description: Blood samples were collected at indicated time points for PK analysis of GSK3739937. PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, 24, 48, 72, 96, 120, 192, 264, and 360 hours post-dose in each treatment period
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 15 | 15
h*ng/mL | 43323.02 (27.3) | 58892.29 (23.6) | 27326.99 (64)
Statistical Analysis 1: Comparison: GSK3739937 Tablet Fed vs GSK3739937 Tablet Fasted; The mixed model was used to estimate Food Effect for the log transformed parameter AUC (0-inf). Analysis was performed using fed/ fasted state and tablet/ PiB as fixed effects and participant as a random effect; Test type: Other; Mixed Models Analysis; Geometric Least Square Mean Ratio = 2.103, 90% CI 2-sided [1.629 to 2.717]
Statistical Analysis 2: Comparison: GSK3739937 PiB Fed vs GSK3739937 Tablet Fed; The mixed model was used to estimate Tablet vs. PiB effect for the log transformed parameter AUC (0-inf). Analysis was performed using the independent variables included a fixed effect for treatment (PiB or Tablet) and period, and participant as a random effect; Test type: Other; Mixed Models Analysis; Geometric Least Square Mean Ratio = 1.351, 90% CI 2-sided [1.22 to 1.497]

72. Primary Outcome: Part 3 - Maximum Observed Concentration (Cmax) of GSK3739937
Description: as for outcome 71
Time Frame: as for outcome 71
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millilitre (ng/mL)
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 16 | 15
nanogram per millilitre (ng/mL) | 389.81 (23.4) | 524.99 (31.8) | 227.88 (93.5)
Statistical Analysis 1: Comparison: GSK3739937 Tablet Fed vs GSK3739937 Tablet Fasted; The mixed model was used to estimate Food Effect for the log transformed parameter Cmax. Analysis was performed using fed/ fasted state and tablet/ PiB as fixed effects and participant as a random effect; Test type: Other; Mixed Models Analysis; Geometric Least Square Mean Ratio = 2.307, 90% CI 2-sided [1.668 to 3.19]
Statistical Analysis 2: Comparison: GSK3739937 PiB Fed vs GSK3739937 Tablet Fed; The mixed model was used to estimate Tablet vs. PiB effect for the log transformed parameter Cmax. Analysis was performed using the independent variables included a fixed effect for treatment (PiB or Tablet) and period, and participant as a random effect; Test type: Other; Mixed Models Analysis; Geometric Least Square Mean Ratio = 1.372, 90% CI 2-sided [1.19 to 1.582]

73. Secondary Outcome: Part 1 (Cohort 1 and 2) - AUC(0-24) of GSK3739937
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12 and 24 hours post-dose in each treatment period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL | 637.8486 (38.8) | 1976.944 (24.3) | 5027.183 (27.4) | 9490.296 (15.4) | 13743.02 (23.6) | 23829.99 (53.1) | 42129.36 (18.1)

74. Secondary Outcome: Part 1 (Cohort 1 and 2) - AUC From Zero (Pre-dose) to Time of the Last Quantifiable Concentration (t) (AUC [0-t]) of GSK3739937
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 12, 24, 48, 72, 96, 120, 192, 264 and 360 hours post-dose in each treatment period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
h*ng/mL | 2486.061 (46.4) | 11441.28 (31.5) | 33650.11 (42.5) | 64937.76 (18.4) | 90730.34 (25.9) | 158068.4 (70) | 293636.9 (33.6)

75. Secondary Outcome: Part 1 (Cohort 1 and 2) - AUC(0-inf) of GSK3739937
Description: as for outcome 71
Time Frame: as for outcome 74
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 5 | 3 | 6
h*ng/mL | NA (NA) — 'NA' refers to not quantifiable as the GSK3739937 concentration was below the lower limit of quantification (10 ng/mL) | 12788.34 (32.4) | 40287.05 (15.5) | 75181.6 (13.6) | 107211.7 (25.2) | 190803.9 (81.6) | 302147.5 (34.2)

76. Secondary Outcome: Part 1 (Cohort 1 and 2) - Apparent Terminal Phase Half-life (T1/2) of GSK3739937
Description: as for outcome 71
Time Frame: as for outcome 74
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 5 | 3 | 6
Hours | NA (NA) — 'NA' refers to not quantifiable as the GSK3739937 concentration was below the lower limit of quantification (10 ng/mL) | 75.8706 (7.4) | 79.0711 (14.4) | 91.8314 (13.6) | 96.7684 (22.7) | 82.6113 (9) | 67.4404 (9.3)

77. Secondary Outcome: Part 1 (Cohort 1 and 2) - Apparent Oral Clearance (CL/F) of GSK3739937
Description: as for outcome 71
Time Frame: as for outcome 74
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: litre/ hour (L/h)
Arm/Group | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 6 | 5 | 4 | 5 | 5 | 3 | 6
litre/ hour (L/h) | NA (NA) — 'NA' refers to not quantifiable as the GSK3739937 concentration was below the lower limit of quantification (10 ng/mL) | 2.3459 (32.4) | 1.9857 (15.5) | 2.1282 (13.6) | 2.9847 (25.2) | 3.3542 (81.6) | 2.6477 (34.2)

78. Secondary Outcome: Part 1 (Cohort 1 and 2) - Cmax of GSK3739937
Description: as for outcome 71
Time Frame: as for outcome 74
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 39.22 (41.6) | 127.3 (22.9) | 310.43 (21) | 528.63 (13.5) | 1014.31 (30.7) | 1458.44 (52) | 2863.33 (22.2)

79. Secondary Outcome: Part 1 (Cohort 1 and 2) - Concentration of GSK3739937 at 24 Hours (C24) of GSK3739937
Description: as for outcome 71
Time Frame: Pre-dose, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 12, 16 and 24 hours post-dose in each treatment period
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 29.46 (37.9) | 85.3 (25.9) | 247.73 (40) | 429.55 (19.4) | 612.15 (14.6) | 1126.32 (71.1) | 2645.7 (31.9)

80. Secondary Outcome: Part 1 (Cohort 1 and 2) - Last Quantifiable Concentration (Clast) of GSK3739937
Description: as for outcome 71
Time Frame: as for outcome 74
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 15.09 (31.1) | 14.41 (23.7) | 18.24 (54.1) | 39.54 (38.7) | 51.33 (70.4) | 78.7 (72.8) | 83.43 (58.1)

81. Secondary Outcome: Part 1 (Cohort 1 and 2 ) - Time of Occurrence of Cmax (Tmax) of GSK3739937
Description: as for outcome 71
Time Frame: as for outcome 74
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours | 6.98 [6 to 8] | 8 [5 to 12.1] | 7.98 [5 to 24.1] | 7.95 [7.95 to 24] | 6.99 [6 to 8] | 7 [5 to 24.2] | 18.08 [12.1 to 24.1]

82. Secondary Outcome: Part 1 (Cohort 1 and 2) - Lag Time (Tlag) of GSK3739937
Description: as for outcome 71
Time Frame: as for outcome 74
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours | 3.47 [2.5 to 4.6] | 1.99 [1.5 to 3] | 1.23 [0.9 to 2] | 1 [0.5 to 1.5] | 1 [0 to 1.1] | 0.5 [0 to 1] | 0 [0 to 1]

83. Secondary Outcome: Part 1 (Cohort 1 and 2) - Time to Reach Clast (Tlast) of GSK3739937
Description: as for outcome 71
Time Frame: as for outcome 74
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6
Hours | 95.7 [95.55 to 192.15] | 261.967 [192.07 to 287.8] | 359.967 [263.38 to 383.82] | 358.942 [335.88 to 363.72] | 359.642 [359.23 to 360.62] | 359.9 [336.27 to 430.33] | 360.334 [358.93 to 362.85]

84. Secondary Outcome: Part 2 (Cohort 3, 4 and 5) - AUC (0-24) of GSK3739937 on Day 1
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 7 | 7 | 7
h*ng/mL | 1888.173 (24.6) | 3559.102 (26.3) | 5893.917 (54.8)

85. Secondary Outcome: Part 2 (Cohort 3, 4 and 5) - Cmax of GSK3739937 on Day 1
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 7 | 7 | 7
ng/mL | 132.12 (23.3) | 232.07 (30) | 375.26 (50.2)

86. Secondary Outcome: Part 2 (Cohort 3, 4 and 5) - C24 of GSK3739937 on Day 1
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 7 | 7 | 7
ng/mL | 89.33 (26.9) | 188.65 (41.1) | 271.59 (75.3)

87. Secondary Outcome: Part 2 (Cohort 3, 4 and 5) - Tmax of GSK3739937 on Day 1
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 1
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 7 | 7 | 7
Hours | 9 [6 to 16] | 8 [7 to 23.8] | 9 [6 to 23.8]

88. Secondary Outcome: Part 2 (Cohort 3, 4 and 5) - Tlag of GSK3739937 on Day 1
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 1
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg
Number analyzed (Participants) | 7 | 7 | 7
Hours | 2 [1 to 4] | 2 [1 to 2] | 1.03 [0.9 to 2.0]

89. Secondary Outcome: Part 2 (Cohort 3 and 4) - Tmax of GSK3739937 on Day 14
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 14
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hour
Arm/Group | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg
Number analyzed (Participants) | 7 | 7
Hour | 6.95 [0 to 9] | 7.03 [3 to 9]

90. Secondary Outcome: Part 2 (Cohort 3 and 4) - Cmax of GSK3739937 on Day 14
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 14
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg
Number analyzed (Participants) | 7 | 7
ng/mL | 766.32 (16) | 1149.32 (15.1)

91. Secondary Outcome: Part 2 (Cohort 3 and 4) - AUC From Pre-dose to the End of the Dosing Interval at Steady State (AUC[0-tau]) of GSK3739937 on Day 14
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 14
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg
Number analyzed (Participants) | 7 | 7
h*ng/mL | 14592.19 (12.6) | 24888.49 (14.4)

92. Secondary Outcome: Part 2 (Cohort 3 and 4) - Plasma Trough Concentration (Ctau) of GSK3739937 on Day 14
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 14
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg
Number analyzed (Participants) | 7 | 7
ng/mL | 588.1557 (22.5) | 990.3205 (13.2)

93. Secondary Outcome: Part 2 (Cohort 3 and 4) - T1/2 of GSK3739937 on Day 14
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 14
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg
Number analyzed (Participants) | 3 | 6
Hours | 85.7725 (25.9) | 72.2484 (28.4)

94. Secondary Outcome: Part 2 (Cohort 3 and 4) - CL/F of GSK3739937 on Day 14
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 14
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg
Number analyzed (Participants) | 7 | 7
L/h | 1.7132 (12.6) | 2.009 (14.4)

95. Secondary Outcome: Part 2 (Cohort 5) - Tmax of GSK3739937 on Day 18
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 18
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3739937 QD 100 mg
Number analyzed (Participants) | 6
Hours | 9.01 [8.1 to 24.1]

96. Secondary Outcome: Part 2 (Cohort 5) - Cmax of GSK3739937 on Day 18
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 18
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3739937 QD 100 mg
Number analyzed (Participants) | 6
ng/mL | 2748 (21.1)

97. Secondary Outcome: Part 2 (Cohort 5) - AUC From Pre-dose to the End of the Dosing Interval at Steady State (AUC[0-tau]) on Day 18
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 18
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | GSK3739937 QD 100 mg
Number analyzed (Participants) | 6
h*ng/mL | 58417.64 (21)

98. Secondary Outcome: Part 2 (Cohort 5) - Plasma Trough Concentration (Ctau) of GSK3739937 on Day 18
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 18
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3739937 QD 100 mg
Number analyzed (Participants) | 6
ng/mL | 2458.275 (21.2)

99. Secondary Outcome: Part 2 (Cohort 5) - T1/2 of GSK3739937 on Day 18
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 18
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | GSK3739937 QD 100 mg
Number analyzed (Participants) | 6
Hours | 78.5264 (26.7)

100. Secondary Outcome: Part 2 (Cohort 5) - CL/F of GSK3739937 on Day 18
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 18
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre/ hour (L/h)
Arm/Group | GSK3739937 QD 100 mg
Number analyzed (Participants) | 6
Litre/ hour (L/h) | 1.7118 (21)

101. Secondary Outcome: Part 2 (Cohort 6) - AUC From Zero to 168 Hours (AUC[0-168]) of GSK3739937 From Day 1
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and up to 168 hours post-dose from Day 1
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | GSK3739937 QW 500 mg
Number analyzed (Participants) | 7
h*ng/mL | 96434.63 (14.1)

102. Secondary Outcome: Part 2 (Cohort 6) - Cmax of GSK3739937 on Day 1
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3739937 QW 500 mg
Number analyzed (Participants) | 7
ng/mL | 1106.61 (12.8)

103. Secondary Outcome: Part 2 (Cohort 6) - Concentration of GSK3739937 at 168 Hours (C168) From Day 1
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and up to 168 hours post-dose from Day 1
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3739937 QW 500 mg
Number analyzed (Participants) | 7
ng/mL | 250.62 (36.3)

104. Secondary Outcome: Part 2 (Cohort 6) - Tmax of GSK3739937 on Day 1
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 1
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3739937 QW 500 mg
Number analyzed (Participants) | 7
Hours | 9.88 [8 to 48.1]

105. Secondary Outcome: Part 2 (Cohort 6) - Tlag of GSK3739937 on Day 1
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 1
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3739937 QW 500 mg
Number analyzed (Participants) | 7
Hours | 0 [0 to 1]

106. Secondary Outcome: Part 2 (Cohort 6 ) - AUC(0-t) of GSK3739937 on Day 15
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 15
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | GSK3739937 QW 500 mg
Number analyzed (Participants) | 7
h*ng/mL | 169693.1 (31.9)

107. Secondary Outcome: Part 2 (Cohort 6) - Cmax of GSK3739937 on Day 15
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 15
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3739937 QW 500 mg
Number analyzed (Participants) | 7
ng/mL | 1855.67 (24.1)

108. Secondary Outcome: Part 2 (Cohort 6) - Ctau of GSK3739937 on Day 15
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 15
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3739937 QW 500 mg
Number analyzed (Participants) | 7
ng/mL | 455.4447 (46.5)

109. Secondary Outcome: Part 2 (Cohort 6) - Tmax of GSK3739937 on Day 15
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 15
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3739937 QW 500 mg
Number analyzed (Participants) | 7
Hours | 10 [9 to 12]

110. Secondary Outcome: Part 2 (Cohort 6) - T1/2 of GSK3739937 on Day 15
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 15
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | GSK3739937 QW 500 mg
Number analyzed (Participants) | 7
Hours | 74.5404 (19.1)

111. Secondary Outcome: Part 2 (Cohort 6) - CL/F of GSK3739937 on Day 15
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on Day 15
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | GSK3739937 QW 500 mg
Number analyzed (Participants) | 7
L/h | 2.9465 (31.9)

112. Secondary Outcome: Part 3 (Cohort 7) - C24 of GSK3739937
Description: as for outcome 71
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16, 24 hours post-dose in each treatment period
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- GSK3739937 Tablet Fasted: In Cohort 7 of Part 3, participants received single oral dose of 100 mg of GSK3739937 Tablet under moderate fasted conditions in each one of the three periods.
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 16 | 15
ng/mL | 316.7 (29.4) | 407.5 (39.7) | 153.97 (91.2)

113. Secondary Outcome: Part 3 (Cohort 7) Clast of GSK3739937
Description: as for outcome 71
Time Frame: as for outcome 71
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 16 | 15
ng/mL | 19.76 (40.8) | 25.09 (51.6) | 15.44 (37)

114. Secondary Outcome: Part 3 (Cohort 7) - Tmax of GSK3739937
Description: as for outcome 71
Time Frame: as for outcome 71
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 16 | 15
Hours | 9 [7 to 24] | 8.42 [5 to 15.9] | 6 [4 to 47.7]

115. Secondary Outcome: Part 3 (Cohort 7) - Tlag of GSK3739937
Description: as for outcome 71
Time Frame: as for outcome 71
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 16 | 15
Hours | 1 [0 to 2] | 2 [0 to 3] | 0.98 [0 to 3]

116. Secondary Outcome: Part 3 (Cohort 7) - Tlast of GSK3739937
Description: as for outcome 71
Time Frame: as for outcome 71
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 15 | 16 | 15
Hours | 336.75 [263.63 to 389.92] | 360.067 [120.08 to 362.27] | 267.4 [195.12 to 361.15]

117. Secondary Outcome: Part 3 (Cohort 7) - T1/2 of GSK3739937
Description: as for outcome 71
Time Frame: as for outcome 71
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 13 | 15 | 10
Hours | 74.7429 (21.5) | 72.9842 (17.5) | 72.8066 (16.9)

118. Secondary Outcome: Part 3 (Cohort 7) - CL/F of GSK3739937
Description: as for outcome 71
Time Frame: as for outcome 71
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
Number analyzed (Participants) | 13 | 15 | 10
L/h | 2.3082 (27.3) | 1.698 (23.6) | 3.6594 (64)

119. Secondary Outcome: Part 1 - Dose Proportionality of GSK3739937 for Dose Levels 30 mg to 800 mg Using AUC(0-infinity) After Single Dose Administration of GSK3739937
Description: Blood samples were collected at indicated time points for PK analysis of GSK3739937. PK parameters were analyzed using standard non-compartmental analysis. Dose proportionality for dose 30 mg, 80 mg, 160 mg, 320 mg, 640 mg and 800 mg was assessed using Power model. Log-e(dose) was fitted as fixed effect and participant was fitted as random effect. Kenward and Roger method and unstructured covariance structure was used. Slope and 90% confidence interval (CI) for the slope are presented.
Time Frame: Up to day 16
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Groups:
- Part 1: GSK3739937 Single Dose of 30 mg to 800 mg: Participants received single dose of GSK3739937 30 mg, 80 mg, 160 mg, 320 mg, 640 mg and 800 mg in either of treatment Period 1, 2 and 3 according to randomization schedule.
Arm/Group | Part 1: GSK3739937 Single Dose of 30 mg to 800 mg
Number analyzed (Participants) | 28
Slope of log dose | 0.882 [0.784 to 0.976]

120. Secondary Outcome: Part 1 - Dose Proportionality of GSK3739937 for Dose Levels 10 mg to 800 mg Using Cmax After Single Dose Administration of GSK3739937
Description: Blood samples were collected at indicated time points for PK analysis of GSK3739937. PK parameters were analyzed using standard non-compartmental analysis. Dose proportionality for dose 10 mg, 30 mg, 80 mg, 160 mg, 320 mg, 640 mg and 800 mg was assessed using Power model. Log-e(dose) was fitted as fixed effect and participant was fitted as random effect. Kenward and Roger method and unstructured covariance structure was used. Slope and 90% confidence interval (CI) for the slope are presented.
Time Frame: Up to day 16
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Groups:
- Part 1: GSK3739937 Single Dose of 10 mg to 800 mg: Participants received single dose of GSK3739937 10 mg, 30 mg, 80 mg, 160 mg, 320 mg, 640 mg and 800 mg in either of treatment Period 1, 2, and 3 according to randomization schedule.
Arm/Group | Part 1: GSK3739937 Single Dose of 10 mg to 800 mg
Number analyzed (Participants) | 42
Slope of log dose | 0.914 [0.855 to 0.966]

121. Secondary Outcome: Part 2 - Dose Proportionality of GSK3739937 for Dose Levels 25 mg to 100 mg Using AUC(0-24) After Repeated Dose Administration of GSK3739937
Description: Blood samples were collected at indicated time points for PK analysis of GSK3739937. PK parameters were analyzed using standard non-compartmental analysis. Dose proportionality for dose 25 mg, 50 mg and 100 mg was assessed using Power model. Log-e(dose) was fitted as fixed effect and participant was fitted as random effect. Kenward and Roger method and unstructured covariance structure was used. Slope and 90% confidence interval (CI) for the slope are presented.
Time Frame: Up to day 33
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Groups:
- Part 2: GSK3739937 Repeated Dose of 25 mg to 100 mg: Participants received repeated dose of GSK3739937 25 mg, 50 mg and 100 mg in treatment Period 1.
Arm/Group | Part 2: GSK3739937 Repeated Dose of 25 mg to 100 mg
Number analyzed (Participants) | 21
Slope of log dose | 0.997 [0.864 to 1.109]

122. Secondary Outcome: Part 2 - Dose Proportionality of GSK3739937 for Dose Levels 25 mg to 100 mg Using Cmax After Repeated Dose Administration of GSK3739937
Description: as for outcome 121
Time Frame: Up to day 33
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Arm/Group | Part 2: GSK3739937 Repeated Dose of 25 mg to 100 mg
Number analyzed (Participants) | 28
Slope of log dose | 0.914 [0.777 to 1.066]

123. Secondary Outcome: Part 2 - Dose Proportionality of GSK3739937 for Dose Levels 25 mg to 100 mg Using Ctau After Repeated Dose Administration of GSK3739937
Description: as for outcome 121
Time Frame: Up to day 33
Population: Pharmacokinetic Population. Only those participants with data available at specified time points have been analyzed.
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Arm/Group | Part 2: GSK3739937 Repeated Dose of 25 mg to 100 mg
Number analyzed (Participants) | 27
Slope of log dose | 1.023 [0.878 to 1.184]

124. Secondary Outcome: Part 2 (Cohort 3 and 4) - Accumulation Ratio of AUC(0-tau) (R [AUC{0-TAU}])
Description: Blood samples were collected at indicated time points for PK analysis of GSK3739937. PK parameters were analyzed using standard non-compartmental analysis. Accumulation ratio calculated as the ratio of day 14 AUC(0-tau) / day 1 AUC(0-tau).
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on both Day 1 and Day 14
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg
Number analyzed (Participants) | 7 | 7
Ratio | 7.728 [6.418 to 9.305] | 6.993 [6.025 to 8.117]

125. Secondary Outcome: Part 2 (Cohort 5) - Accumulation Ratio of AUC(0-tau) (R [AUC{0-TAU}])
Description: Blood samples were collected at indicated time points for PK analysis of GSK3739937. PK parameters were analyzed using standard non-compartmental analysis. Accumulation ratio calculated as the ratio of day 18 AUC(0-tau) / day 1 AUC(0-tau).
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on both Day 1 and Day 18
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | GSK3739937 QD 100 mg
Number analyzed (Participants) | 7
Ratio | 9.943 [6.987 to 14.149]

126. Secondary Outcome: Part 2 (Cohort 6) - Accumulation Ratio of AUC(0-tau) (R [AUC{0-TAU}])
Description: Blood samples were collected at indicated time points for PK analysis of GSK3739937. PK parameters were analyzed using standard non-compartmental analysis. Accumulation ratio calculated as the ratio of day 15 AUC(0-tau) / day 1 AUC(0-tau).
Time Frame: Pre-dose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 and 16 hours post-dose on both Day 1 and Day 15
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | GSK3739937 QW 500 mg
Number analyzed (Participants) | 7
Ratio | 1.76 [1.448 to 2.138]

127. Secondary Outcome: Part 2 (Cohort 3 and 4) - Accumulation Ratio of Cmax (R [CMAX])
Description: Blood samples were collected at indicated time points for PK analysis of GSK3739937. PK parameters were analyzed using standard non-compartmental analysis. Accumulation ratio calculated as the ratio of day 14 Cmax / day 1 Cmax.
Time Frame: as for outcome 124
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg
Number analyzed (Participants) | 7 | 7
Ratio | 5.8 [4.962 to 6.78] | 4.952 [4.198 to 5.842]

128. Secondary Outcome: Part 2 (Cohort 5) - Accumulation Ratio of Cmax (R [CMAX])
Description: Blood samples were collected at indicated time points for PK analysis of GSK3739937. PK parameters were analyzed using standard non-compartmental analysis. Actual measure type is Ratio. Accumulation ratio calculated as the ratio of day 18 Cmax / day 1 Cmax.
Time Frame: as for outcome 125
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | GSK3739937 QD 100 mg
Number analyzed (Participants) | 7
Ratio | 7.325 [5.333 to 10.06]

129. Secondary Outcome: Part 2 (Cohort 6) - Accumulation Ratio of Cmax (R [CMAX])
Description: Blood samples were collected at indicated time points for PK analysis of GSK3739937. PK parameters were analyzed using standard non-compartmental analysis. Accumulation ratio calculated as the ratio of day 15 Cmax / day 1 Cmax.
Time Frame: as for outcome 126
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | GSK3739937 QW 500 mg
Number analyzed (Participants) | 7
Ratio | 1.677 [1.381 to 2.036]

130. Secondary Outcome: Part 2 (Cohort 3 and 4) - Accumulation Ratio of C(Tau) (R[CTAU])
Description: Blood samples were collected at indicated time points for PK analysis of GSK3739937. PK parameters were analyzed using standard non-compartmental analysis. Accumulation ratio calculated as the ratio of day 14 C(Tau) / day 1 C(Tau).
Time Frame: as for outcome 124
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg
Number analyzed (Participants) | 7 | 7
Ratio | 6.584 [5.256 to 8.248] | 5.25 [4.07 to 6.771]

131. Secondary Outcome: Part 2 (Cohort 5) - Accumulation Ratio of C(Tau) (R[CTAU])
Description: Blood samples were collected at indicated time points for PK analysis of GSK3739937. PK parameters were analyzed using standard non-compartmental analysis. Accumulation ratio calculated as the ratio of day 18 C(Tau) / day 1 C(Tau).
Time Frame: as for outcome 125
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | GSK3739937 QD 100 mg
Number analyzed (Participants) | 7
Ratio | 9.133 [5.562 to 14.995]

132. Secondary Outcome: Part 2 (Cohort 6) - Accumulation Ratio of C(Tau) (R[CTAU])
Description: Blood samples were collected at indicated time points for PK analysis of GSK3739937. PK parameters were analyzed using standard non-compartmental analysis. Accumulation ratio calculated as the ratio of day 15 C(Tau) / day 1 C(Tau).
Time Frame: as for outcome 126
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Ratio
Arm/Group | GSK3739937 QW 500 mg
Number analyzed (Participants) | 7
Ratio | 1.817 [1.428 to 2.313]

133. Secondary Outcome: Part 2 (Cohort 3 and 4) - Pre-dose Concentration of GSK3739937
Description: Blood samples were collected at indicated time points for PK analysis of GSK3739937. For Part 2 cohorts 3 and 4, steady-state GSK3739937 concentrations was assessed by estimating the slope of concentrations on pre-dose assessments on Days 2-14 (Part 2 cohort 3 and 4) and the day 15 (24-hr post-dose relative to dosing on day 14). PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Up to day 15
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Arm/Group | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg
Number analyzed (Participants) | 7 | 7
Slope of log dose | 37.1872 [33.0332 to 41.3412] | 57.1056 [51.9304 to 62.2808]

134. Secondary Outcome: Part 2 (Cohort 5) - Pre-dose Concentration of GSK3739937
Description: Blood samples were collected at indicated time points for PK analysis of GSK3739937. For Part 2 cohort 5, steady state GSK3739937 concentrations was assessed by estimating the slope of the concentrations of pre-dose assessments on Days 2-18 and the day 19 (24-hr post-dose relative to dosing on day 18). PK parameters were analyzed using standard non-compartmental analysis.
Time Frame: Up to day 19
Population: Pharmacokinetic Population
Measure: Number (90% Confidence Interval); unit: Slope of log dose
Arm/Group | GSK3739937 QD 100 mg
Number analyzed (Participants) | 7
Slope of log dose | 114.9742 [103.8293 to 126.119]

ADVERSE EVENTS:
Time Frame: All cause mortality, Non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to 27 weeks in Part 1, up to 5 weeks in Part 2 and up to 16 weeks in Part 3.
Description: Safety population included all randomized participants who received at least one dose of study treatment. Data is presented treatment-wise.
Arm/Group | Placebo (PBO) Single Dose | GSK3739937 Single Dose (SD) 10 mg | GSK3739937 SD 30 mg | GSK3739937 SD 80 mg | GSK3739937 SD 160 mg | GSK3739937 SD 320 mg | GSK3739937 SD 640 mg | GSK3739937 SD 800 mg | PBO Once Daily (QD) | GSK3739937 QD 25 mg | GSK3739937 QD 50 mg | GSK3739937 QD 100 mg | PBO Once Weekly (QW) | GSK3739937 QW 500 mg | GSK3739937 PiB Fed | GSK3739937 Tablet Fed | GSK3739937 Tablet Fasted
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/7 | 0/7 | 0/7 | 0/3 | 0/7 | 0/15 | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/9 | 0/7 | 0/7 | 0/7 | 0/3 | 0/7 | 0/15 | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 4/21 | 1/6 | 3/6 | 3/6 | 0/6 | 2/6 | 4/6 | 2/6 | 3/9 | 0/7 | 2/7 | 5/7 | 0/3 | 4/7 | 2/15 | 4/17 | 6/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (PBO) Single Dose (N=21) | GSK3739937 Single Dose (SD) 10 mg (N=6) | GSK3739937 SD 30 mg (N=6) | GSK3739937 SD 80 mg (N=6) | GSK3739937 SD 160 mg (N=6) | GSK3739937 SD 320 mg (N=6) | GSK3739937 SD 640 mg (N=6) | GSK3739937 SD 800 mg (N=6) | PBO Once Daily (QD) (N=9) | GSK3739937 QD 25 mg (N=7) | GSK3739937 QD 50 mg (N=7) | GSK3739937 QD 100 mg (N=7) | PBO Once Weekly (QW) (N=3) | GSK3739937 QW 500 mg (N=7) | GSK3739937 PiB Fed (N=15) | GSK3739937 Tablet Fed (N=17) | GSK3739937 Tablet Fasted (N=15)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site dermatitis (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Burn oral cavity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premenstrual pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT04493684/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT04493684/SAP_001.pdf